CLINICAL TRIAL: NCT00205777
Title: Fracture Incidence Reduction And Safety Of TSE-424 (Bazedoxifene Acetate) Compared To Placebo And Raloxifene In Osteoporotic Postmenopausal Women
Brief Title: Study Evaluating Bazedoxifene Acetate In Osteoporosis In Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3068A1-301; B1781001
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Results first posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-02

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Postmenopause
MeSH Terms: conditions — Osteoporosis | interventions — bazedoxifene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Bazedoxifene Acetate
- B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bazedoxifene Acetate — BZA 20mg, daily, oral
  Arms: A
Other: Placebo — Placebo, daily, oral
  Arms: B

SUMMARY:
The purpose of this study is to determine whether bazedoxifene acetate is safe and effective in the treatment of osteoporosis in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 2 years postmenopausal
* Osteoporotic subjects without vertebral fracture who meet BMD criteria, or Osteoporotic subjects with vertebral fracture

Exclusion Criteria:

* Diseases that may affect bone metabolism
* Vasomotor symptoms requiring treatment
* Known history or suspected cancer of the breast
* Active or past history of venous thromboembolic events

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7609 (Actual)
Dates: Start 2001-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (257):
- United States (144):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, Palm Desert, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Rancho Mirage, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, Bridgeport, Connecticut
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, Madison, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Cape Coral, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Delray Beach, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Holiday, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Largo, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Port Orange, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Riverdale, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Cadwell, Idaho
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Meridian, Idaho
  - Pfizer Investigational Site, Champaign, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Libertyville, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Avon, Indiana
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Lousiville, Kentucky
  - Pfizer Investigational Site, Bangor, Maine
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Silver Spring, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Brookline, Massachusetts
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Kalamazaoo, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Brooklyn Center, Minnesota
  - Pfizer Investigational Site, Robbinsdale, Minnesota
  - Pfizer Investigational Site, Shoreview, Minnesota
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Bozeman, Montana
  - Pfizer Investigational Site, Missoula, Montana
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, North Las Vegas, Nevada
  - Pfizer Investigational Site, Reno, Nevada
  - Pfizer Investigational Site, Manchester Twp, New Jersey
  - Pfizer Investigational Site, Ocean City, New Jersey
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Jamestown, North Dakota
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Oakes, North Dakota
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Centerville, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Lyndhurst, Ohio
  - Pfizer Investigational Site, Mayfield Village, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Yukon, Oklahoma
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Camp Hill, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Langhome, Pennsylvania
  - Pfizer Investigational Site, Lemoyne, Pennsylvania
  - Pfizer Investigational Site, Newtown, Pennsylvania
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Belton, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Aberdeen, South Dakota
  - Pfizer Investigational Site, Sioux Falls, South Dakota
  - Pfizer Investigational Site, Waterdown, South Dakota
  - Pfizer Investigational Site, Watertown, South Dakota
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Bellaire, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Waco, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, Cheyenne, Wyoming
- Pfizer Investigational Site, Provincia de Buenos Aires, Argentina
- Australia (5):
  - Pfizer Investigational Site, Concord, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Nedlands, Western Australia
  - Pfizer Investigational Site, Herston
  - Pfizer Investigational Site, Keswick
- Pfizer Investigational Site, Graz, Austria
- Belgium (6):
  - Pfizer Investigational Site, Ghent, Belgium
  - Pfizer Investigational Site, Liège, Liege
  - Pfizer Investigational Site, Diepenbeek
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Schiepsebos
- Brazil (5):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Duque de Caxias - Cuiaba, Mato Grosso
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, São Paulo, São Paulo
  - Pfizer Investigational Site, Sorocaba, São Paulo
- Bulgaria (5):
  - Pfizer Investigational Site, Plovdiv, Bulgaria
  - Pfizer Investigational Site, Sofia, Bulgaria
  - Pfizer Investigational Site, Pleven
  - Pfizer Investigational Site, Plovdiv
  - Pfizer Investigational Site, Sofia
- Canada (14):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Gatineau, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Trois-Rivières, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Pfizer Investigational Site, Santiago, Chile
- Croatia (2):
  - Pfizer Investigational Site, Zadar
  - Pfizer Investigational Site, Zagreb
- Denmark (3):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Ballerup Municipality
  - Pfizer Investigational Site, Vejle
- Estonia (2):
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- Finland (6):
  - Pfizer Investigational Site, Oulu, Finland
  - Pfizer Investigational Site, Jyväskylä, FIN
  - Pfizer Investigational Site, Jyväskylä
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Lahti
  - Pfizer Investigational Site, Turku
- France (3):
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Orléans
  - Pfizer Investigational Site, Paris
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Zerbst
- Pfizer Investigational Site, Athens, Greece, Greece
- Hong Kong (3):
  - Pfizer Investigational Site, Hong Kong
  - Pfizer Investigational Site, PRC
  - Pfizer Investigational Site, Sai Ying Pung
- Hungary (4):
  - Pfizer Investigational Site, Békéscsaba
  - Pfizer Investigational Site, H-6720 Szeged
  - Pfizer Investigational Site, Kecskemét
  - Pfizer Investigational Site, Makó
- Italy (2):
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Siena
- Lithuania (2):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Vilnius
- Mexico (2):
  - Pfizer Investigational Site, Seccion de Lomas Verdes, State of Mexico
  - Pfizer Investigational Site, Mexico City
- Netherlands (6):
  - Pfizer Investigational Site, Emmen, Drenthe
  - Pfizer Investigational Site, Nijmegen, GA
  - Pfizer Investigational Site, Amsterdam, HV
  - Pfizer Investigational Site, Nijmegen, SZ
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Rotterdam
- New Zealand (4):
  - Pfizer Investigational Site, Milford, Auckland
  - Pfizer Investigational Site, Christchurch, NZ
  - Pfizer Investigational Site, Auckland
  - Pfizer Investigational Site, Dunedin
- Norway (4):
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Hamar
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Trondheim
- Poland (7):
  - Pfizer Investigational Site, Krakow, Krakow
  - Pfizer Investigational Site, Katowice, Poland
  - Pfizer Investigational Site, Warsaw, Poland
  - Pfizer Investigational Site, Wroclaw, Poland
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Warsaw
- Romania (5):
  - Pfizer Investigational Site, Iași, Iaşi
  - Pfizer Investigational Site, Cluj-Napoca, Napoca
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Bucharesti
  - Pfizer Investigational Site, Cluj-Napoca
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Slovakia (2):
  - Pfizer Investigational Site, Piešťany, Slovak Republic
  - Pfizer Investigational Site, Bratislava
- South Africa (9):
  - Pfizer Investigational Site, Groenkloof, Pretoria
  - Pfizer Investigational Site, Johannesburg, South Africa
  - Pfizer Investigational Site, Pretoria, South Africa
  - Pfizer Investigational Site, Bedford Gardens
  - Pfizer Investigational Site, Johannesburg
  - Pfizer Investigational Site, Parow
  - Pfizer Investigational Site, Pretoria
  - Pfizer Investigational Site, Somerset West
  - Pfizer Investigational Site, Stellenbosch
- Spain (3):
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Madrid, Spain
  - Pfizer Investigational Site, Madrid

REFERENCES:
- [Derived] Christiansen C, Chesnut CH 3rd, Adachi JD, Brown JP, Fernandes CE, Kung AW, Palacios S, Levine AB, Chines AA, Constantine GD. Safety of bazedoxifene in a randomized, double-blind, placebo- and active-controlled Phase 3 study of postmenopausal women with osteoporosis. BMC Musculoskelet Disord. 2010 Jun 22;11:130. doi: 10.1186/1471-2474-11-130. PMID 20569451
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3068A1-301&StudyName=Study%20Evaluating%20Bazedoxifene%20Acetate%20In%20Osteoporosis%20In%20Postmenopausal%20Women

RESULTS

PARTICIPANT FLOW:
Groups:
- Bazedoxifene 20 mg (Core+SE I): Bazedoxifene acetate 20 milligram (mg) capsule orally once daily for 3 years in the core study and further 2 years in study extension I (SE I), along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 international unit [IU]) orally twice daily.
- Bazedoxifene 40 mg (Core): Bazedoxifene acetate 40 mg capsule orally once daily for 3 years in the core study, along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily.
- Raloxifene 60 mg (Core): Raloxifene 60 mg capsule orally once daily for 3 years in the core study, along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily.
- Placebo (Core+SE I+SE II): Matching placebo capsule orally once daily for 3 years in the core study, further 2 years in study extension I (SE I) and further 2 years in study extension II (SE II), along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily.
- Bazedoxifene 40/20 mg (SE I): Participants from Bazedoxifene 40 mg treatment arm continued to receive bazedoxifene acetate 40 mg capsule orally once daily in first year of study extension I and then dose reduced to bazedoxifene acetate 20 mg in second year of study extension I, along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily.
- Bazedoxifene 20 mg (SE II): Participants from Bazedoxifene 20 mg and Bazedoxifene 40/20 mg treatment arm received bazedoxifene 20 mg capsule orally once daily for further 2 years in study extension II, along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily.
Period: Core Study (Up to 3 Years)
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I) | Bazedoxifene 20 mg (SE II)
Started | 1907 | 1904 | 1884 | 1914 | 0 | 0
TREATED | 1886 | 1872 | 1849 | 1885 | 0 | 0
Completed | 1279 | 1245 | 1277 | 1282 | 0 | 0
Not Completed | 628 | 659 | 607 | 632 | 0 | 0
Not completed — Adverse Event | 260 | 267 | 252 | 232 | 0 | 0
Not completed — Death | 9 | 7 | 14 | 7 | 0 | 0
Not completed — Failed to return | 40 | 25 | 27 | 27 | 0 | 0
Not completed — Other Event | 49 | 52 | 41 | 58 | 0 | 0
Not completed — Withdrawal by Subject | 144 | 169 | 149 | 162 | 0 | 0
Not completed — Protocol Violation | 53 | 55 | 50 | 42 | 0 | 0
Not completed — Lack of Efficacy | 52 | 52 | 39 | 75 | 0 | 0
Not completed — Randomized but not treated | 21 | 32 | 35 | 29 | 0 | 0
Period: Completed Core Study, Entered SE I
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I) | Bazedoxifene 20 mg (SE II)
Started | 1279 | 1245 | 1277 | 1282 | 0 | 0
Completed | 1047 | 1041 | 1070 | 1058 | 0 | 0
Not Completed | 232 | 204 | 207 | 224 | 0 | 0
Not completed — Withdrawal by Subject | 180 | 158 | 160 | 174 | 0 | 0
Not completed — Other Event | 52 | 46 | 47 | 50 | 0 | 0
Period: Study Extension I
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I) | Bazedoxifene 20 mg (SE II)
Started | 1047 | 0 | 1070 | 1058 | 1041 | 0
Completed | 833 | 0 | 0 | 830 | 840 | 0
Not Completed | 214 | 0 | 1070 | 228 | 201 | 0
Not completed — Adverse Event | 57 | 0 | 0 | 61 | 58 | 0
Not completed — Death | 5 | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 99 | 0 | 0 | 106 | 89 | 0
Not completed — Protocol Violation | 4 | 0 | 0 | 8 | 8 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Failed to return | 15 | 0 | 0 | 17 | 13 | 0
Not completed — Other Event | 34 | 0 | 0 | 34 | 29 | 0
Not completed — Withdrawn as per protocol | 0 | 0 | 1070 | 0 | 0 | 0
Period: Completed SE I, Entered Extension SE II
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I) | Bazedoxifene 20 mg (SE II)
Started | 833 | 0 | 0 | 830 | 840 | 0
Completed | 560 | 0 | 0 | 590 | 582 | 0
Not Completed | 273 | 0 | 0 | 240 | 258 | 0
Not completed — No-consent/eligible/SEII continuing site | 273 | 0 | 0 | 240 | 258 | 0
Period: Study Extension II
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I) | Bazedoxifene 20 mg (SE II)
Started | 0 | 0 | 0 | 590 | 0 | 1142
TREATED | 0 | 0 | 0 | 519 | 0 | 1011
Completed | 0 | 0 | 0 | 441 | 0 | 860
Not Completed | 0 | 0 | 0 | 149 | 0 | 282
Not completed — Adverse Event | 0 | 0 | 0 | 14 | 0 | 30
Not completed — Death | 0 | 0 | 0 | 2 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 35 | 0 | 59
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 10
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Failed to return | 0 | 0 | 0 | 14 | 0 | 26
Not completed — Other Event | 0 | 0 | 0 | 12 | 0 | 20
Not completed — Enrolled but not treated | 0 | 0 | 0 | 71 | 0 | 131

BASELINE CHARACTERISTICS:
Groups:
- Bazedoxifene 20 mg (Core+SE I): Bazedoxifene acetate 20 mg capsule orally once daily for 3 years in the core study and further 2 years in study extension I (SE I), along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 international unit [IU]) orally twice daily.
- Total: Total of all reporting groups
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II) | Total
Number analyzed (Participants) | 1886 | 1872 | 1849 | 1885 | 7492
Age Continuous [Mean (Standard Deviation); unit: years] | 66.48 (6.53) | 66.22 (6.80) | 66.36 (6.74) | 66.47 (6.76) | 66.38 (6.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1886 | 1872 | 1849 | 1885 | 7492
  Male | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Height (cm) was measured 3 times using standardized Harpenden stadiometer (height based on the middle stadiometer reading was recorded). Number of participants analyzed (N) = 1883, 1869, 1848, 1883 for each arm group.
  centimeter (cm) | 156.60 (7.21) | 156.28 (7.38) | 156.37 (7.23) | 156.35 (6.90) | 156.40 (7.18)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With New Vertebral Fractures Through Month 36
Description: New vertebral fracture: decrease in anterior, mid, or posterior vertebral (vt) height of approximately 20% and 4 millimeter (mm) or more from baseline (base) to end of study confirmed by measurement of involved vt body, a semi-quantitative grade change of 1 from base for any vertebra from fourth thoracic to fourth lumbar vertebra (T4 to L4), provided vertebra was not fractured at base. Participant was counted only once irrespective of how many new vt fractures were diagnosed. Stratification factor was base fracture status, categorized as no prevalent fracture and at least 1 prevalent fracture.
Time Frame: Baseline through Month 36
Population: Intent-to-treat(ITT) population for vt fractures:randomized participants who took at least 1 dose of test article;had vt radiographic assessment at baseline and at least once while on therapy.N (number of participants analyzed)=participants evaluable for this measure.n=participants with specified baseline fracture status evaluable for each group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1724 | 1686 | 1696 | 1741
Percentage of participants
  No Prevalent Fracture (n=757,744,742,760) | 1.98 [1.15 to 3.40] | 2.14 [1.25 to 3.67] | 1.84 [1.04 to 3.22] | 3.13 [2.03 to 4.82]
  At Least 1 Prevalent Fracture (n=967,942,954,981) | 2.63 [1.73 to 3.98] | 2.80 [1.86 to 4.20] | 2.74 [1.81 to 4.14] | 4.80 [3.52 to 6.52]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% confidence intervals (CIs); Test type: Superiority or Other; p = 0.22, Log Rank; Hazard Ratio (HR) = 0.647, 95% CI 2-sided [0.322 to 1.302]
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 40 mg [Core] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.24, Log Rank; Hazard Ratio (HR) = 0.647, 95% CI 2-sided [0.322 to 1.301]
Statistical Analysis 3: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 40 mg [Core] versus Raloxifene 60 mg [Core]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.83, Log Rank; Hazard Ratio (HR) = 1.097, 95% CI 2-sided [0.501 to 2.405]
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Raloxifene 60 mg [Core]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.87, Log Rank; Hazard Ratio (HR) = 1.074, 95% CI 2-sided [0.490 to 2.356]
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40 mg (Core); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Bazedoxifene 40 mg [Core]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.96, Log Rank; Hazard Ratio (HR) = 0.988, 95% CI 2-sided [0.458 to 2.131]
Statistical Analysis 6: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Raloxifene 60 mg [Core] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.16, Log Rank; Hazard Ratio (HR) = 0.592, 95% CI 2-sided [0.289 to 1.212]
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); At Least 1 Prevalent Fracture: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.035, Log Rank; Hazard Ratio (HR) = 0.551, 95% CI 2-sided [0.324 to 0.937]
Statistical Analysis 8: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); At Least 1 Prevalent Fracture: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 40 mg [Core] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.070, Log Rank; Hazard Ratio (HR) = 0.624, 95% CI 2-sided [0.373 to 1.045]
Statistical Analysis 9: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); At Least 1 Prevalent Fracture: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 40 mg [Core] versus Raloxifene 60 mg [Core]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.79, Log Rank; Hazard Ratio (HR) = 1.085, 95% CI 2-sided [0.605 to 1.947]
Statistical Analysis 10: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); At Least 1 Prevalent Fracture: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Raloxifene 60 mg [Core]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.99, Log Rank; Hazard Ratio (HR) = 0.959, 95% CI 2-sided [0.527 to 1.743]
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40 mg (Core); At Least 1 Prevalent Fracture: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Bazedoxifene 40 mg [Core]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.78, Log Rank; Hazard Ratio (HR) = 0.882, 95% CI 2-sided [0.488 to 1.593]
Statistical Analysis 12: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); At Least 1 Prevalent Fracture: P value was calculated using stratified log-rank test. Hazard ratio (Raloxifene 60 mg [Core] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.036, Log Rank; Hazard Ratio (HR) = 0.574, 95% CI 2-sided [0.340 to 0.968]

2. Primary Outcome: Percentage of Participants With New Vertebral Fractures Through Month 60
Description: New vertebral fracture: decrease in anterior, mid, or posterior vt height of approximately 20% and 4 millimeter (mm) or more from baseline (base) to end of study confirmed by measurement of involved vt body, a semi-quantitative grade change of 1 from base for any vertebra from fourth thoracic to fourth lumbar vertebra (T4 to L4), provided vertebra was not fractured at base. Participant was counted only once irrespective of how many new vt fractures were diagnosed. Stratification factor was base fracture status, categorized as no prevalent fracture and at least 1 prevalent fracture.
Time Frame: Baseline through Month 60
Population: ITT population for vt fractures:randomized participants who took at least 1 dose of test article;had vt radiographic assessment at baseline and at least once while on therapy.N (number of participants analyzed)=participants evaluable for this measure.n=participants with specified baseline fracture status evaluable for each group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo (Core+SE I+SE II): Matching placebo capsules orally once daily for 3 years in the core study, further 2 years in study extension I (SE I) and further 2 years in study extension II (SE II), along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily.
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 1724 | 1741 | 1686
Percentage of participants
  No Prevalent Fracture (n=757,760,744) | 3.11 [1.94 to 4.96] | 5.40 [3.73 to 7.80] | 3.46 [2.20 to 5.43]
  At Least 1 Prevalent Fracture (n=967,981,942) | 5.67 [4.05 to 7.92] | 7.95 [6.07 to 10.37] | 4.28 [2.97 to 6.17]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.097, Log Rank; Hazard Ratio (HR) = 0.610, 95% CI 2-sided [0.339 to 1.099]
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 40/20 mg [SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.15, Log Rank; Hazard Ratio (HR) = 0.645, 95% CI 2-sided [0.361 to 1.151]
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40/20 mg (SE I); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Bazedoxifene 40/20 mg [SE I]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.83, Log Rank; Hazard Ratio (HR) = 0.941, 95% CI 2-sided [0.493 to 1.793]
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; p = 0.067, Log Rank; Hazard Ratio (HR) = 0.666, 95% CI 2-sided [0.435 to 1.019]
Statistical Analysis 5: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); At Least 1 Prevalent Fracture: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 40/20 mg [SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.014, Log Rank; Hazard Ratio (HR) = 0.573, 95% CI 2-sided [0.367 to 0.896]
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40/20 mg (SE I); At Least 1 Prevalent Fracture: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Bazedoxifene 40/20 mg [SE I]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.50, Log Rank; Hazard Ratio (HR) = 1.157, 95% CI 2-sided [0.710 to 1.885]

3. Primary Outcome: Percentage of Participants With New Vertebral Fractures Through Month 84
Description: as for outcome 2
Time Frame: Baseline through Month 84
Population: Modified ITT(mITT) population of safety population category one(SP1) population:randomized participants who took at least 1 dose of test article;had vt radiographic assessment at baseline and at least once while on therapy.N (number of participants analyzed)=participants evaluable.n=participants with specified baseline fracture status.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Core+SE I+SE II) | Bazedoxifene 20 mg (SE II)
Number analyzed (Participants) | 1741 | 3410
Percentage of participants
  No Prevalent Fracture (n=760,1501) | 8.18 [5.73 to 11.61] | 5.79 [4.24 to 7.89]
  At Least 1 Prevalent Fracture (n=981,1909) | 11.35 [8.63 to 14.86] | 6.90 [5.32 to 8.92]
Statistical Analysis 1: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); No Prevalent Fractures: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [SE II] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.085, Log Rank; Hazard Ratio (HR) = 0.680, 95% CI 2-sided [0.440 to 1.052]
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); At Least 1 Prevalent Fracture: P value was calculated using stratified log-rank test. Hazard ratio (Bazedoxifene 20 mg [SE II] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.004, Log Rank; Hazard Ratio (HR) = 0.610, 95% CI 2-sided [0.434 to 0.857]

4. Secondary Outcome: Incidence of Breast Cancer Through Month 36
Description: Incidence of breast cancer was defined as the number of participants with breast cancer diagnosis by the time point of interest divided by the number of participants included in the analysis. The reported rate was rescaled to reflect average follow-up time per 1000 women (1000 multiplied by number of cases divided by total follow-up time).
Time Frame: Baseline through Month 36
Population: Safety Population 1 (SP1) included all randomized participants who received at least 1 dose of test article. 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Number; unit: Breast cancer per 1000-women years
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1885 | 1872 | 1849 | 1885
Breast cancer per 1000-women years | 1.09 | 0.90 | 1.55 | 1.74
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); P value was calculated using logistic regression. Gail index was added to the model to account for baseline risk differences between participants; Test type: Superiority or Other; p = 0.40, Regression, Logistic; Odds Ratio (OR) = 0.621, 95% CI 2-sided [0.203 to 1.903]
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.26, Regression, Logistic; Odds Ratio (OR) = 0.504, 95% CI 2-sided [0.151 to 1.676]
Statistical Analysis 3: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.33, Regression, Logistic; Odds Ratio (OR) = 0.540, 95% CI 2-sided [0.157 to 1.860]
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.49, Regression, Logistic; Odds Ratio (OR) = 0.661, 95% CI 2-sided [0.206 to 2.118]
Statistical Analysis 5: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.76, Regression, Logistic; Odds Ratio (OR) = 0.850, 95% CI 2-sided [0.305 to 2.370]
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40 mg (Core); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.75, Regression, Logistic; Odds Ratio (OR) = 1.238, 95% CI 2-sided [0.332 to 4.616]

5. Secondary Outcome: Incidence of Breast Cancer Through Month 60
Description: as for outcome 4
Time Frame: Baseline through Month 60
Population: SP1 included all randomized participants who received at least 1 dose of test article. 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Number; unit: Breast cancer per 1000-women years
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 1885 | 1885 | 1872
Breast cancer per 1000-women years | 1.40 | 1.56 | 1.43
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Relative risk versus placebo was provided together with 95% CIs; Test type: Superiority or Other; Relative Risk = 0.9, 95% CI 2-sided [0.38 to 2.15]
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Relative risk versus placebo was provided together with 95% CIs; Test type: Superiority or Other; Relative Risk = 0.92, 95% CI 2-sided [0.39 to 2.21]

6. Secondary Outcome: Incidence of Breast Cancer Through Month 84
Description: as for outcome 4
Time Frame: Baseline through Month 84
Population: as for outcome 5
Measure: Number; unit: Breast cancer per 1000-women years
Arm/Group | Placebo (Core+SE I+SE II) | Bazedoxifene 20 mg (SE II)
Number analyzed (Participants) | 1885 | 3757
Breast cancer per 1000-women years | 1.50 | 1.52
Statistical Analysis 1: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Relative risk versus placebo was provided together with 95% CIs; Test type: Superiority or Other; Relative risk = 1.01, 95% CI 2-sided [0.5 to 2.06]

7. Secondary Outcome: Percentage of Participants With New Clinical Vertebral Fractures Through Month 36
Description: A new clinical vertebral fracture was defined as a new fracture found at any time because of back pain suggestive of fracture(s). New Clinical vertebral fractures were verified with radiographic assessment using both semi-quantitative and quantitative morphometric assessment: decrease in anterior, mid, or posterior vt height of approximately 20% and 4 mm or more from base to end of study confirmed by measurement of involved vt body, a semi-quantitative grade change of 1 from base for any vertebra from T4 to L4, provided vertebra was not fractured at base.
Time Frame: Baseline through Month 36
Population: ITT population for vt fractures:randomized participants who took at least 1 dose of test article;had vt radiographic assessment at baseline and at least once while on therapy. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1724 | 1686 | 1696 | 1741
Percentage of participants | 0.72 [0.40 to 1.31] | 0.76 [0.42 to 1.37] | 0.87 [0.51 to 1.50] | 0.94 [0.56 to 1.58]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.57, Log Rank
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.62, Log Rank
Statistical Analysis 3: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.72, Log Rank
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.67, Log Rank
Statistical Analysis 5: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.89, Log Rank
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40 mg (Core); Test type: Superiority or Other; p = 0.95, Log Rank

8. Secondary Outcome: Percentage of Participants With New Clinical Vertebral Fractures Through Month 60
Description: as for outcome 7
Time Frame: Baseline through Month 60
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 1724 | 1741 | 1686
Percentage of participants | 0.79 [0.45 to 1.39] | 1.37 [0.85 to 2.21] | 0.84 [0.47 to 1.47]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.29, Log Rank
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.31, Log Rank
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.94, Log Rank

9. Secondary Outcome: Percentage of Participants With New Clinical Vertebral Fractures Through Month 84
Description: as for outcome 7
Time Frame: Baseline through Month 84
Population: mITT population of SP1 population included all randomized participants who took at least 1 dose of test article and who had a vertebral radiographic assessment at baseline and at least once while on therapy. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Core+SE I+SE II) | Bazedoxifene 20 mg (SE II)
Number analyzed (Participants) | 1741 | 3410
Percentage of participants | 1.92 [1.20 to 3.08] | 1.28 [0.82 to 1.97]
Statistical Analysis 1: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Test type: Superiority or Other; p = 0.18, Log Rank

10. Secondary Outcome: Number of Participants With Worsening Vertebral Fractures Through Month 36
Description: A worsening vertebral fracture was defined as a decrease in anterior, mid, or posterior vertebral height of at least 20% and at least 4 mm as evaluated by quantitative morphometric assessment, and a grade change of at least 1 as rated by a radiologist using the semi-quantitative rating scale. It can occur only in a vertebra that was fractured at baseline.
Time Frame: Baseline through Month 36
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1724 | 1686 | 1696 | 1741
Participants | 3 | 2 | 2 | 1

11. Secondary Outcome: Number of Participants With Worsening Vertebral Fractures Through Month 60
Description: as for outcome 10
Time Frame: Baseline through Month 60
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 1724 | 1741 | 1686
Participants | 4 | 1 | 2

12. Secondary Outcome: Number of Participants With Worsening Vertebral Fractures Through Month 84
Description: as for outcome 10
Time Frame: Baseline through Month 84
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Placebo (Core+SE I+SE II) | Bazedoxifene 20 mg (SE II)
Number analyzed (Participants) | 1741 | 3410
Participants | 1 | 7

13. Secondary Outcome: Percentage of Participants With Non-vertebral Fractures Through Month 36
Description: Non-vertebral fractures were determined by direct questioning at each clinic visit after medication therapy begins. Osteoporosis-related, hip and wrist fractures were summarized.
Time Frame: Baseline through Month 36
Population: ITT population for vt fractures:randomized participants who took at least 1 dose of test article;had vt radiographic assessment at baseline and at least once while on therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1886 | 1872 | 1849 | 1885
Percentage of participants
  Osteoporosis-Related | 5.68 [4.63 to 6.96] | 5.61 [4.55 to 6.90] | 5.87 [4.79 to 7.19] | 6.26 [5.16 to 7.59]
  Hip | 0.55 [0.28 to 1.05] | 0.34 [0.14 to 0.82] | 0.26 [0.10 to 0.69] | 0.31 [0.13 to 0.75]
  Wrist | 2.28 [1.63 to 3.18] | 1.83 [1.25 to 2.67] | 2.51 [1.83 to 3.44] | 1.64 [1.12 to 2.41]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Osteoporosis-Related: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.46, Log Rank
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40 mg (Core); Osteoporosis-Related: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.90, Log Rank
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Osteoporosis-Related: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.93, Log Rank
Statistical Analysis 4: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Osteoporosis-Related: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.84, Log Rank
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Osteoporosis-Related: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.39, Log Rank
Statistical Analysis 6: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Osteoporosis-Related: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.52, Log Rank
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Hip: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.28, Log Rank
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40 mg (Core); Hip: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.31, Log Rank
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Hip: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.17, Log Rank
Statistical Analysis 10: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Hip: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.72, Log Rank
Statistical Analysis 11: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Hip: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.97, Log Rank
Statistical Analysis 12: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Hip: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.76, Log Rank
Statistical Analysis 13: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Wrist: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.29, Log Rank
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40 mg (Core); Wrist: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.43, Log Rank
Statistical Analysis 15: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Wrist: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.59, Log Rank
Statistical Analysis 16: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Wrist: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.19, Log Rank
Statistical Analysis 17: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Wrist: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.80, Log Rank
Statistical Analysis 18: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Wrist: P value was calculated using Log-Rank test; Test type: Superiority or Other; p = 0.11, Log Rank

14. Secondary Outcome: Percentage of Participants With Non-vertebral Fractures Through Month 60
Description: as for outcome 13
Time Frame: Baseline through Month 60
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 1886 | 1872 | 1885
Percentage of participants
  Osteoporosis-Related | 9.47 [7.96 to 11.25] | 9.03 [7.58 to 10.74] | 7.59 [6.27 to 9.18]
  Hip | 0.75 [0.41 to 1.38] | 0.65 [0.31 to 1.33] | 0.53 [0.25 to 1.12]
  Wrist | 3.30 [2.45 to 4.45] | 2.79 [2.01 to 3.88] | 2.60 [1.85 to 3.66]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Osteoporosis-Related: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.968, Log Rank; Hazard Ratio (HR) = 1.012, 95% CI 2-sided [0.790 to 1.296]
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Osteoporosis-Related: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 40/20 mg [SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.211, Log Rank; Hazard Ratio (HR) = 0.846, 95% CI 2-sided [0.652 to 1.097]
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40/20 mg (SE I); Osteoporosis-Related: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Bazedoxifene 40/20 mg [SE I]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.191, Log Rank; Hazard Ratio (HR) = 1.200, 95% CI 2-sided [0.925 to 1.556]
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Hip: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.493, Log Rank; Hazard Ratio (HR) = 1.406, 95% CI 2-sided [0.566 to 3.497]
Statistical Analysis 5: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Hip: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 40/20 mg [SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.820, Log Rank; Hazard Ratio (HR) = 0.872, 95% CI 2-sided [0.316 to 2.405]
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40/20 mg (SE I); Hip: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Bazedoxifene 40/20 mg [SE I]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.371, Log Rank; Hazard Ratio (HR) = 1.612, 95% CI 2-sided [0.624 to 4.161]
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Wrist: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.423, Log Rank; Hazard Ratio (HR) = 1.202, 95% CI 2-sided [0.776 to 1.861]
Statistical Analysis 8: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Wrist: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 40/20 mg [SE I] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.799, Log Rank; Hazard Ratio (HR) = 0.936, 95% CI 2-sided [0.587 to 1.491]
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40/20 mg (SE I); Wrist: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 20 mg [Core+SE I] versus Bazedoxifene 40/20 mg [SE I]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.298, Log Rank; Hazard Ratio (HR) = 1.280, 95% CI 2-sided [0.818 to 2.002]

15. Secondary Outcome: Percentage of Participants With Non-vertebral Fractures Through Month 84
Description: as for outcome 13
Time Frame: Baseline through Month 84
Population: mITT population of SP1 population:randomized participants who took at least 1 dose of test article;had vt radiographic assessment at baseline and at least once while on therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Core+SE I+SE II) | Bazedoxifene 20 mg (SE II)
Number analyzed (Participants) | 1885 | 3758
Percentage of participants
  Osteoporosis-Related | 10.77 [8.98 to 12.89] | 11.20 [9.79 to 12.79]
  Hip | 1.34 [0.68 to 2.63] | 0.74 [0.46 to 1.21]
  Wrist | 3.62 [2.59 to 5.07] | 4.61 [3.66 to 5.79]
Statistical Analysis 1: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Osteoporosis-Related: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 20 mg [SE II] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.73, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.78 to 1.19]
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Hip: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 20 mg [SE II] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.71, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.41 to 1.83]
Statistical Analysis 3: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Wrist: P value was calculated using Log-Rank test. Hazard ratio (Bazedoxifene 20 mg [SE II] versus Placebo [Core+SE I+SE II]) based on a Cox proportional hazards regression model was presented along with 95% CIs; Test type: Superiority or Other; p = 0.45, Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.80 to 1.66]

16. Secondary Outcome: Change From Baseline in Height at Month 36
Description: Height was measured 3 times using standardized Harpenden stadiometer (height based on the middle stadiometer reading was recorded).
Time Frame: Baseline, Month 36
Population: ITT population for vt fractures:randomized participants who took at least 1 dose of test article;had vt radiographic assessment at baseline and at least once while on therapy. N (number of participants analyzed)=participants evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1236 | 1210 | 1231 | 1254
millimeter (mm) | -3.7 (0.31) | -3.9 (0.31) | -4.5 (0.31) | -3.3 (0.31)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.31, ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.039, ANCOVA
Statistical Analysis 3: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.13, ANCOVA
Statistical Analysis 4: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.12, ANCOVA
Statistical Analysis 5: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.002, ANCOVA

17. Secondary Outcome: Change From Baseline in Height at Month 60
Description: as for outcome 16
Time Frame: Baseline, Month 60
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 746 | 752 | 743
mm | -0.50 (0.06) | -0.41 (0.06) | -0.41 (0.06)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.12, ANCOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.94, ANCOVA

18. Secondary Outcome: Change From Baseline in Height at Month 84
Description: Height (cm) was measured 3 times using standardized Harpenden stadiometer (height based on the middle stadiometer reading was recorded).
Time Frame: Baseline, Month 84
Population: mITT population of SP1 population:randomized participants who took at least 1 dose of test article;had vt radiographic assessment at baseline and at least once while on therapy. 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo (Core+SE I+SE II) | Bazedoxifene 20 mg (SE II)
Number analyzed (Participants) | 407 | 736
mm | -0.68 (0.10) | -0.73 (0.08)
Statistical Analysis 1: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Test type: Superiority or Other; p = 0.26, ANCOVA

19. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at Month 6, 12, 18, 24 and 36
Description: BMD of lumbar spine (Lu Sp) and hip (total hip [Tl Hp], femoral neck [Fe Ne] and femur trochanter [Fe Tr]) was evaluated by dual-energy x-ray absorptiometry (DXA). The left hip was evaluated unless prevented by pathology, in which case the right hip was evaluated throughout the study. Results were scored as T score, defined as BMD at the site when compared to the young normal reference mean. Normal BMD is a T-score of -1.0 or higher.
Time Frame: Baseline, Months 6, 12, 18, 24, 36
Population: ITT population included all randomized participants who took at least 1 dose of test article; had baseline BMD and at least one valid BMD while on therapy. N (number of participants analyzed)=participants evaluable for this measure.n=participants with specified baseline fracture status evaluable for each group.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1693 | 1663 | 1662 | 1711
Percent change
  Lu Sp:Change at Month 6 (n=1693,1663,1662,1711) | 1.53 (0.09) | 1.56 (0.09) | 1.79 (0.09) | 0.51 (0.09)
  Tl Hp:Change at Month 6 (n=1684,1653,1659,1699) | 0.75 (0.07) | 0.85 (0.07) | 1.07 (0.07) | 0.24 (0.06)
  Fe Ne:Change at Month 6 (n=1687,1658,1662,1703) | 0.60 (0.09) | 0.62 (0.09) | 0.52 (0.09) | -0.05 (0.09)
  Fe Tr:Change at Month 6 (n=1687,1658,1662,1703) | 1.17 (0.10) | 1.24 (0.10) | 1.49 (0.10) | 0.33 (0.10)
  Lu Sp:Change at Month 12 (n=1587,1541,1546,1599) | 2.06 (0.10) | 2.13 (0.10) | 2.50 (0.10) | 0.61 (0.10)
  Tl Hp:Change at Month 12 (n=1578,1532,1532,1586) | 1.07 (0.07) | 1.24 (0.08) | 1.50 (0.08) | 0.28 (0.07)
  Fe Ne:Change at Month 12 (n=1581,1537,1536,1591) | 0.92 (0.09) | 1.10 (0.10) | 1.27 (0.10) | 0.08 (0.09)
  Fe Tr:Change at Month 12 (n=1581,1537,1536,1591) | 1.71 (0.11) | 1.84 (0.11) | 2.14 (0.11) | 0.63 (0.11)
  Lu Sp:Change at Month 18 (n=1498,1444,1474,1487) | 2.00 (0.11) | 2.24 (0.11) | 2.58 (0.11) | 0.52 (0.11)
  Tl Hp:Change at Month 18 (n=1486,1434,1459,1480) | 0.93 (0.08) | 1.13 (0.08) | 1.47 (0.08) | -0.07 (0.08)
  Fe Ne:Change at Month 18 (n=1489,1437,1463,1484) | 0.80 (0.10) | 1.09 (0.10) | 1.21 (0.10) | -0.24 (0.10)
  Fe Tr:Change at Month 18 (n=1489,1437,1463,1484) | 1.54 (0.12) | 1.64 (0.12) | 2.18 (0.12) | 0.14 (0.12)
  Lu Sp:Change at Month 24 (n=1400,1347,1387,1398) | 1.99 (0.11) | 2.12 (0.11) | 2.74 (0.11) | 0.47 (0.11)
  Tl Hp:Change at Month 24 (n=1394,1333,1379,1382) | 0.82 (0.09) | 1.01 (0.09) | 1.37 (0.09) | -0.35 (0.09)
  Fe Ne:Change at Month 24 (n=1398,1335,1381,1386) | 0.80 (0.10) | 1.05 (0.11) | 1.37 (0.10) | -0.58 (0.10)
  Fe Tr:Change at Month 24 (n=1398,1335,1381,1386) | 1.51 (0.12) | 1.57 (0.13) | 2.18 (0.13) | 0.01 (0.13)
  Lu Sp:Change at Month 36 (n=1022,1029,1050,1054) | 2.21 (0.16) | 2.38 (0.16) | 2.96 (0.16) | 0.88 (0.16)
  Tl Hp:Change at Month 36 (n=1019,1016,1044,1050) | 0.27 (0.12) | 0.50 (0.12) | 0.90 (0.12) | -0.83 (0.12)
  Fe Ne:Change at Month 36 (n=1020,1018,1046,1051) | 0.28 (0.15) | 0.67 (0.15) | 0.80 (0.15) | -1.30 (0.15)
  Fe Tr:Change at Month 36 (n=1020,1018,1046,1051) | 0.89 (0.17) | 0.90 (0.17) | 1.62 (0.17) | -0.50 (0.17)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in lumbar spine BMD: P value was calculated using Analysis of covariance (ANCOVA); Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.018, ANCOVA
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 18 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 10: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 11: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 12: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 13: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 14: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 15: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 16: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.036, ANCOVA
Statistical Analysis 17: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.003, ANCOVA
Statistical Analysis 18: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 18 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.019, ANCOVA
Statistical Analysis 19: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 20: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.002, ANCOVA
Statistical Analysis 21: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 22: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 23: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 24: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 25: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 26: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 27: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 28: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 29: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 30: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 31: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 32: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 33: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 18 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 34: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 35: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 36: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 37: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 38: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 39: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 40: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 41: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.008, ANCOVA
Statistical Analysis 42: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.007, ANCOVA
Statistical Analysis 43: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 18 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.002, ANCOVA
Statistical Analysis 44: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.002, ANCOVA
Statistical Analysis 45: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.006, ANCOVA
Statistical Analysis 46: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 47: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 48: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 49: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 50: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 51: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 52: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 53: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 54: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 55: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 56: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.47, ANCOVA
Statistical Analysis 57: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.005, ANCOVA
Statistical Analysis 58: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 18 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.002, ANCOVA
Statistical Analysis 59: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 60: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.004, ANCOVA
Statistical Analysis 61: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 62: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 63: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 64: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 65: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 66: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.39, ANCOVA
Statistical Analysis 67: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.17, ANCOVA
Statistical Analysis 68: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 18 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.34, ANCOVA
Statistical Analysis 69: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.016, ANCOVA
Statistical Analysis 70: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.47, ANCOVA
Statistical Analysis 71: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 72: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 73: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 74: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 75: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 76: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 77: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 78: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 79: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 80: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 81: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.01, ANCOVA
Statistical Analysis 82: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.002, ANCOVA
Statistical Analysis 83: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 18 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 84: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 85: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 86: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 87: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 88: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 89: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 90: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 91: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.048, ANCOVA
Statistical Analysis 92: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.038, ANCOVA
Statistical Analysis 93: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 18 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 94: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 95: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 96: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 97: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 98: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 18 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 99: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 100: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA

20. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at Months 48, 60
Description: as for outcome 19
Time Frame: Baseline, Month 48, 60
Population: mITT population of SP1 population:randomized participants who took at least 1 dose of test article; had baseline BMD and at least one valid BMD while on therapy. N (number of participants analyzed)=participants evaluable for this measure.n=participants with specified baseline fracture status evaluable for each group.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 886 | 876 | 886
Percent change
  Lu Sp:Change at Month 48 (n=886,876,886) | 1.92 (0.22) | 0.84 (0.22) | 2.02 (0.22)
  Tl Hp:Change at Month 48 (n=877,865,868) | -0.17 (0.18) | -1.05 (0.18) | 0.11 (0.18)
  Fe Ne:Change at Month 48 (n=879,866,870) | 0.02 (0.20) | -1.30 (0.20) | 0.45 (0.20)
  Fe Tr:Change at Month 48 (n=879,734,870) | 0.18 (0.24) | -0.81 (0.25) | 0.45 (0.25)
  Lu Sp:Change at Month 60 (n=742,747,746) | 2.16 (0.26) | 1.46 (0.26) | 2.08 (0.26)
  Tl Hp:Change at Month 60 (n=738,733,736) | -0.48 (0.21) | -1.49 (0.21) | -0.29 (0.21)
  Fe Ne:Change at Month 60 (n=740,734,737) | -0.18 (0.25) | -1.72 (0.25) | 0.09 (0.25)
  Fe Tr:Change at Month 60 (n= 740,734,737) | -0.13 (0.29) | -1.19 (0.29) | -0.00 (0.29)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 48 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 60 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.010, ANCOVA
Statistical Analysis 3: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 48 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 60 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.023, ANCOVA
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 48 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 60 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 48 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 60 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 48 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 10: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 60 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 11: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 48 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 12: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 60 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 13: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 48 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 60 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 15: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 48 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 16: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 60 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA

21. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at Months 72 and 84
Description: as for outcome 19
Time Frame: Baseline, Month 72, 84
Population: Modified ITT(mITT) population of SP1 population:randomized participants who took at least 1 dose of test article;had baseline BMD and at least one valid BMD while on therapy. N (number of participants analyzed)=participants evaluable.n=participants with specified baseline fracture status.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo (Core+SE I+SE II) | Bazedoxifene 20 mg (SE II)
Number analyzed (Participants) | 457 | 888
Percent change
  Lu Sp:Change at Month 72 (n=457,888) | 1.80 (0.40) | 2.24 (0.31)
  Tl Hp:Change at Month 72 (n=448,871) | -1.96 (0.33) | -0.85 (0.25)
  Fe Ne:Change at Month 72 (n=448,871) | -2.12 (0.39) | -0.60 (0.30)
  Fe Tr:Change at Month 72 (n=448,871) | -1.43 (0.44) | -0.31 (0.34)
  Lu Sp:Change at Month 84 (n=417,800) | 2.19 (0.49) | 2.95 (0.39)
  Tl Hp:Change at Month 84 (n=405,787) | -2.53 (0.38) | -1.15 (0.30)
  Fe Ne:Change at Month 84 (n=405,787) | -2.35 (0.43) | -0.80 (0.35)
  Fe Tr:Change at Month 84 (n=405,787) | -2.72 (0.47) | -1.41 (0.38)
Statistical Analysis 1: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 72 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.34, ANCOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 84 in lumbar spine BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.15, ANCOVA
Statistical Analysis 3: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 72 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 84 in total hip BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 72 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 84 in femoral neck BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 72 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.003, ANCOVA
Statistical Analysis 8: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 84 in femoral trochanter BMD: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.002, ANCOVA

22. Secondary Outcome: Percent Change From Baseline in Osteocalcin at Month 3, 6 and 12
Description: Osteocalcin is a biochemical marker of bone formation. Blood samples were collected to evaluate osteocalcin levels.
Time Frame: Baseline, Months 3, 6, 12
Population: ITT population included all randomized participants who took at least 1 dose of test article. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' is signifying those participants who were evaluable for this measure at the specified time point for each arm group.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1739 | 1708 | 1702 | 1746
Percent change
  Change at Month 3 (n=1739,1708,1702,1746) | -23.48 [-33.69 to -10.56] | -25.28 [-35.72 to -14.50] | -26.18 [-36.33 to -13.95] | -11.37 [-22.75 to 1.60]
  Change at Month 6 (n=1655,1634,1633,1681) | -32.75 [-44.07 to -19.01] | -35.20 [-46.05 to -22.77] | -35.96 [-45.91 to -23.67] | -17.82 [-30.48 to -3.82]
  Change at Month 12 (n=1565,1522,1529,1573) | -37.49 [-48.43 to -22.09] | -39.15 [-51.16 to -25.78] | -41.44 [-51.98 to -28.78] | -21.00 [-34.41 to -4.52]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 3 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 3 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 3: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 3 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 4: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 3 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.93, Ranked ANCOVA
Statistical Analysis 5: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 3 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 8: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 9: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.30, Ranked ANCOVA
Statistical Analysis 10: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 12: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 13: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 14: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 15: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA

23. Secondary Outcome: Percent Change From Baseline in Osteocalcin at Months 36 and 60
Description: Osteocalcin is a biochemical marker of bone formation. Blood samples were collected to evaluate osteocalcin levels.
Time Frame: Baseline, Months 36, 60
Population: mITT of SP1 population included all randomized participants who took at least 1 dose of test article.'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' is signifying those participants who were evaluable for this measure at the specified time point for each arm group.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 178 | 168 | 181
Percent change
  Change at Month 36 (n=178,168,181) | -23.91 [-36.90 to -0.95] | -12.73 [-26.68 to 12.57] | -26.99 [-40.13 to -8.52]
  Change at Month 60 (n=127, 127, 132) | -25.21 [-39.80 to -8.59] | -17.21 [-32.49 to 0.04] | -30.41 [-45.36 to -16.12]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 60 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 3: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 36 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 4: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 60 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA

24. Secondary Outcome: Percent Change From Baseline in Osteocalcin at Months 72 and 84
Description: Osteocalcin is a biochemical marker of bone formation. Blood samples were collected to evaluate osteocalcin levels.
Time Frame: Baseline, Months 72, 84
Population: mITT of SP1 population included all randomized participants who took at least 1 dose of test article. 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo (Core+SE I+SE II) | Bazedoxifene 20 mg (SE II)
Number analyzed (Participants) | 97 | 170
Percent change
  Change at Month 72 (n=97,170) | -26.72 [-43.48 to -9.53] | -33.76 [-49.30 to -13.30]
  Change at Month 84 (n=84,147) | -29.50 [-42.38 to -12.01] | -32.25 [-51.48 to -13.60]
Statistical Analysis 1: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 72 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.037, Ranked ANCOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 84 in osteocalcin: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.16, Ranked ANCOVA

25. Secondary Outcome: Percent Change From Baseline in C-telopeptide (CTx) at Month 3, 6 and 12
Description: C-telopeptide is a biochemical marker of bone formation. Blood samples were collected to evaluate C-telopeptide levels.
Time Frame: Baseline, Months 3, 6, 12
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1739 | 1708 | 1703 | 1746
Percent change
  Change at Month 3 (n=1739,1708,1703,1746) | -42.12 [-57.23 to -23.43] | -45.11 [-60.12 to -27.75] | -45.48 [-60.98 to -28.13] | -26.17 [-44.03 to -5.46]
  Change at Month 6 (n=1655,1634,1634,1681) | -46.93 [-62.75 to -28.18] | -50.00 [-64.99 to -31.42] | -52.55 [-67.27 to -34.00] | -27.94 [-46.27 to -6.65]
  Change at Month 12 (n=1565,1522,1530,1573) | -45.64 [-61.77 to -26.05] | -48.77 [-63.73 to -28.83] | -54.55 [-67.72 to -35.84] | -27.31 [-46.64 to -5.12]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 3 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 3 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 3: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 3 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 4: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 3 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.40, Ranked ANCOVA
Statistical Analysis 5: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 3 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 8: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 9: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.004, Ranked ANCOVA
Statistical Analysis 10: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 12: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 13: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 14: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 15: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA

26. Secondary Outcome: Percent Change From Baseline in C-telopeptide (CTx) at Months 36 and 60
Description: C-telopeptide is a biochemical marker of bone formation. Blood samples were collected to evaluate C-telopeptide levels.
Time Frame: Baseline, Months 36, 60
Population: mITT of SP1 population included all randomized participants who took at least 1 dose of test article. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' is signifying those participants who were evaluable for this measure at the specified time point for each arm group.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 178 | 180 | 168
Percent change
  Change at Month 36 (n=178,180,168) | -30.54 [-46.98 to -10.57] | -21.85 [-37.38 to 3.95] | -32.26 [-51.31 to -11.96]
  Change at Month 60 (n=127,131,126) | -26.80 [-44.82 to 2.47] | -10.40 [-36.16 to 12.82] | -27.87 [-47.58 to 1.97]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 60 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.001, Ranked ANCOVA
Statistical Analysis 3: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 36 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA
Statistical Analysis 4: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Percent change at Month 60 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.009, Ranked ANCOVA

27. Secondary Outcome: Percent Change From Baseline in C-telopeptide (CTx) at Months 72 and 84
Description: C-telopeptide is a biochemical marker of bone formation. Blood samples were collected to evaluate C-telopeptide levels.
Time Frame: Baseline, Months 72, 84
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo (Core+SE I+SE II) | Bazedoxifene 20 mg (SE II)
Number analyzed (Participants) | 97 | 170
Percent change
  Change at Month 72 (n=97,170) | -29.44 [-49.83 to 4.04] | -37.41 [-59.11 to -11.36]
  Change at Month 84 (n=84,147) | -28.61 [-49.04 to 3.92] | -28.17 [-48.02 to 1.70]
Statistical Analysis 1: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 72 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.034, Ranked ANCOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 20 mg (SE II); Percent change at Month 84 in C-telopeptide: P value was calculated using Ranked ANCOVA; Test type: Superiority or Other; p = 0.77, Ranked ANCOVA

28. Secondary Outcome: Percent Change From Baseline in Lipid Parameters at Months 6, 12, 24 and 36
Description: Lipid parameters evaluated included total cholesterol (TC), low density lipoprotein (LDL), high density lipoprotein (HDL), triglyceride (TG), high-density lipoprotein fraction 2 (HDL2) and high-density lipoprotein fraction 3 (HDL3).
Time Frame: Baseline, Months 6, 12, 24, 36
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1647 | 1623 | 1628 | 1674
Percent change
  TC:Change at Month 6 (n=1646,1623,1628,1673) | -3.89 [-11.89 to 4.90] | -4.73 [-12.94 to 4.74] | -5.50 [-13.49 to 3.20] | 0.00 [-8.05 to 9.72]
  LDL:Change at Month 6 (n=1647,1623,1627,1674) | -8.55 [-19.92 to 1.89] | -10.18 [-20.56 to 0.93] | -11.52 [-21.49 to -1.22] | -1.17 [-12.68 to 10.12]
  HDL:Change at Month 6 (n=1647,1619,1626,1671) | 1.43 [-7.19 to 11.39] | 1.06 [-8.09 to 11.81] | 0.00 [-9.15 to 10.71] | 0.00 [-9.46 to 10.00]
  HDL2:Change at Month 6 (n=1643,1618,1623,1666) | -13.89 [-35.21 to 14.63] | -11.86 [-36.00 to 18.18] | -14.75 [-36.11 to 10.20] | -12.22 [-35.71 to 17.11]
  HDL3:Change at Month 6 (n=1643,1619,1625,1668) | 9.38 [-3.41 to 23.68] | 8.60 [-4.50 to 23.08] | 8.70 [-4.35 to 23.08] | 6.90 [-7.14 to 21.01]
  TG:Change at Month 6 (n=1646,1623,1628,1673) | 4.28 [-17.17 to 31.58] | 7.14 [-15.57 to 34.82] | 5.71 [-17.36 to 33.89] | 4.90 [-16.99 to 31.58]
  TC:Change at Month 12 (n=1556,1515,1536,1578) | -4.14 [-12.02 to 4.76] | -3.66 [-11.95 to 4.90] | -5.18 [-12.84 to 2.90] | 0.87 [-6.91 to 9.25]
  LDL:Change at Month 12 (n=1559,1516,1534,1578) | -7.79 [-18.27 to 3.31] | -8.45 [-18.59 to 2.94] | -10.28 [-19.71 to 0.00] | 0.66 [-9.49 to 11.32]
  HDL:Change at Month 12 (n=1552,1513,1531,1576) | 1.14 [-7.78 to 10.24] | 0.66 [-8.60 to 10.75] | 0.58 [-8.39 to 9.26] | -1.17 [-9.57 to 8.63]
  HDL2:Change at Month 12 (n=1550,1510,1528,1570) | -16.55 [-35.71 to 9.52] | -16.33 [-39.74 to 9.62] | -17.54 [-37.34 to 7.32] | -14.29 [-36.47 to 12.82]
  HDL3:Change at Month 12 (n=1551,1511,1531,1572) | 9.85 [-2.15 to 23.81] | 10.00 [-2.63 to 23.81] | 9.52 [-2.13 to 22.86] | 6.38 [-6.67 to 20.00]
  TG:Change at Month 12 (n=1556,1515,1535,1578) | 5.95 [-15.08 to 32.44] | 8.14 [-14.67 to 38.36] | 6.25 [-15.12 to 34.07] | 7.99 [-13.54 to 36.18]
  TC:Change at Month 24 (n=1378,1341,1377,1385) | -4.17 [-12.50 to 6.18] | -4.72 [-12.63 to 4.61] | -5.68 [-13.22 to 2.96] | 0.38 [-8.15 to 9.57]
  LDL:Change at Month 24 (n=1379,1341,1376,1384) | -4.51 [-16.18 to 10.03] | -5.94 [-17.81 to 7.57] | -7.30 [-18.13 to 5.09] | 4.41 [-9.05 to 16.00]
  HDL:Change at Month 24 (n=1377,1338,1374,1382) | 3.57 [-6.25 to 13.50] | 2.42 [-6.74 to 13.16] | 2.41 [-6.74 to 13.37] | 1.63 [-7.55 to 11.68]
  HDL2:Change at Month 24 (n=1369,1336,1363,1377) | -10.26 [-32.81 to 14.29] | -11.94 [-33.87 to 13.00] | -13.04 [-32.69 to 13.46] | -10.61 [-33.33 to 17.07]
  HDL3:Change at Month 24 (n=1370,1337,1365,1379) | 10.81 [-2.17 to 25.24] | 10.77 [-2.15 to 26.39] | 10.99 [-2.27 to 25.27] | 6.98 [-5.38 to 22.22]
  TG:Change at Month 24 (n=1378,1341,1377,1385) | 4.23 [-17.91 to 31.25] | 8.09 [-16.22 to 34.95] | 5.17 [-17.91 to 35.19] | 6.19 [-15.79 to 34.55]
  TC:Change at Month 36 (n=1220,1201,1225,1248) | -3.75 [-11.68 to 5.00] | -3.47 [-12.71 to 5.72] | -5.04 [-13.16 to 3.96] | 0.34 [-8.23 to 9.60]
  LDL:Change at Month 36 (n=1220,1201,1223,1247) | -5.36 [-17.11 to 7.13] | -6.63 [-18.70 to 5.96] | -8.51 [-19.76 to 4.20] | 1.55 [-11.41 to 15.56]
  HDL:Change at Month 36 (n=1216,1196,1219,1246) | 5.10 [-4.33 to 15.56] | 5.93 [-4.23 to 17.01] | 5.00 [-4.91 to 15.33] | 2.51 [-7.59 to 12.57]
  HDL2:Change at Month 36 (n=1209,1191,1214,1236) | -19.51 [-39.22 to 6.12] | -17.07 [-39.29 to 8.89] | -18.47 [-39.22 to 6.82] | -18.66 [-38.10 to 5.56]
  HDL3:Change at Month 36 (n=1210,1194,1218,1237) | 18.18 [3.33 to 32.50] | 17.93 [4.76 to 33.33] | 17.14 [4.39 to 32.56] | 13.33 [0.00 to 28.85]
  TG:Change at Month 36 (n=1220,1201,1225,1248) | 8.48 [-14.97 to 42.26] | 13.59 [-13.70 to 46.91] | 12.21 [-11.65 to 43.66] | 12.11 [-13.53 to 48.62]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 9: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 10: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 11: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 12: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 13: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.009, ANCOVA
Statistical Analysis 14: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 15: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.055, ANCOVA
Statistical Analysis 16: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.004, ANCOVA
Statistical Analysis 17: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 18: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 19: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 20: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in total cholesterol: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 21: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 22: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 23: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 24: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 25: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 26: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 27: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 28: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 29: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 30: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 31: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 32: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 33: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.012, ANCOVA
Statistical Analysis 34: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 35: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.031, ANCOVA
Statistical Analysis 36: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.008, ANCOVA
Statistical Analysis 37: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 38: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 39: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 40: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in LDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 41: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 42: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 43: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 44: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 45: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.10, ANCOVA
Statistical Analysis 46: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.89, ANCOVA
Statistical Analysis 47: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.60, ANCOVA
Statistical Analysis 48: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.82, ANCOVA
Statistical Analysis 49: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 50: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 51: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.012, ANCOVA
Statistical Analysis 52: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 53: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.083, ANCOVA
Statistical Analysis 54: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.96, ANCOVA
Statistical Analysis 55: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.84, ANCOVA
Statistical Analysis 56: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.15, ANCOVA
Statistical Analysis 57: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.13, ANCOVA
Statistical Analysis 58: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 59: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.007, ANCOVA
Statistical Analysis 60: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in HDL: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 61: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.28, ANCOVA
Statistical Analysis 62: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.10, ANCOVA
Statistical Analysis 63: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.94, ANCOVA
Statistical Analysis 64: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.46, ANCOVA
Statistical Analysis 65: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.63, ANCOVA
Statistical Analysis 66: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.70, ANCOVA
Statistical Analysis 67: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.58, ANCOVA
Statistical Analysis 68: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.29, ANCOVA
Statistical Analysis 69: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.59, ANCOVA
Statistical Analysis 70: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.036, ANCOVA
Statistical Analysis 71: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.57, ANCOVA
Statistical Analysis 72: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.49, ANCOVA
Statistical Analysis 73: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.038, ANCOVA
Statistical Analysis 74: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.93, ANCOVA
Statistical Analysis 75: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.96, ANCOVA
Statistical Analysis 76: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.72, ANCOVA
Statistical Analysis 77: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.12, ANCOVA
Statistical Analysis 78: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.043, ANCOVA
Statistical Analysis 79: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.53, ANCOVA
Statistical Analysis 80: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in HDL2: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.75, ANCOVA
Statistical Analysis 81: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 82: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 83: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 84: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 85: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.46, ANCOVA
Statistical Analysis 86: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.64, ANCOVA
Statistical Analysis 87: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.47, ANCOVA
Statistical Analysis 88: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.75, ANCOVA
Statistical Analysis 89: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.003, ANCOVA
Statistical Analysis 90: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 91: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 92: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 93: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.81, ANCOVA
Statistical Analysis 94: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.98, ANCOVA
Statistical Analysis 95: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.87, ANCOVA
Statistical Analysis 96: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.40, ANCOVA
Statistical Analysis 97: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 98: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 99: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 100: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in HDL3: P value was calculated using ANCOVA; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 101: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.85, ANCOVA
Statistical Analysis 102: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.26, ANCOVA
Statistical Analysis 103: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.33, ANCOVA
Statistical Analysis 104: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.22, ANCOVA
Statistical Analysis 105: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 6 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.86, ANCOVA
Statistical Analysis 106: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 12 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.65, ANCOVA
Statistical Analysis 107: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 24 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 1.00, ANCOVA
Statistical Analysis 108: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Percent change at Month 36 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.44, ANCOVA
Statistical Analysis 109: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.058, ANCOVA
Statistical Analysis 110: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.55, ANCOVA
Statistical Analysis 111: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.34, ANCOVA
Statistical Analysis 112: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.96, ANCOVA
Statistical Analysis 113: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 6 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.058, ANCOVA
Statistical Analysis 114: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 12 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.031, ANCOVA
Statistical Analysis 115: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 24 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.054, ANCOVA
Statistical Analysis 116: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Percent change at Month 36 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.62, ANCOVA
Statistical Analysis 117: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 6 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.99, ANCOVA
Statistical Analysis 118: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 12 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.11, ANCOVA
Statistical Analysis 119: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 24 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.33, ANCOVA
Statistical Analysis 120: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Percent change at Month 36 in Triglycerides: P value was calculated using ANCOVA; Test type: Superiority or Other; p = 0.65, ANCOVA

29. Secondary Outcome: Bone Histomorphometric Indices at Month 36: BV, OV, OS, OcS, ObS, MS, ES, OMS, CP
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD. Percentage of following indices (volume,surface,porosity) was calculated:Bone Volume(BV), Osteoid Volume(OV), Osteoid Surface(OS), Osteoclast Surface(OcS), Osteoblast Surface(ObS), Mineralizing surface(MS), Eroded Surface(ES), Osteoid Mineralizing surface(OMS), Cortical porosity(CP).
Time Frame: Month 36
Population: ITT population included all randomized participants who took at least 1 dose of test article; had baseline data and at least one valid bone histomorphometry while on therapy. 'N' (number of participants analyzed)=participants evaluable for this measure. 'n'=participants evaluable for this measure at the specified time point for each arm group.
Measure: Least Squares Mean (Standard Error); unit: Percentage of indices
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 28 | 29 | 32 | 32
Percentage of indices
  BV (n=25,27,28,30) | 17.078 (1.140) | 19.155 (1.097) | 16.650 (1.077) | 17.144 (1.041)
  OV (n=25,27,28,30) | 1.513 (0.244) | 1.644 (0.234) | 1.290 (0.230) | 1.605 (0.222)
  OS (n=25,27,28,30) | 12.516 (1.795) | 14.196 (1.728) | 12.442 (1.697) | 12.934 (1.639)
  OcS (n=25,27,28,30) | 0.276 (0.045) | 0.334 (0.043) | 0.215 (0.043) | 0.242 (0.041)
  ObS (n=25,27,28,30) | 4.235 (0.623) | 4.225 (0.600) | 2.772 (0.589) | 3.672 (0.569)
  MS (n=25,27,28,30) | 5.962 (0.852) | 5.960 (0.820) | 3.926 (0.805) | 5.705 (0.778)
  ES (n=25,27,28,30) | 1.610 (0.196) | 1.855 (0.189) | 1.891 (0.185) | 1.299 (0.179)
  OMS (n=28,29,32,32) | 49.629 (5.442) | 49.145 (5.347) | 37.856 (5.091) | 51.503 (5.091)
  CP (n=25,27,27,29) | 4.484 (0.397) | 4.130 (0.382) | 4.319 (0.382) | 4.334 (0.369)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); BV: P value was calculated using Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.97, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); BV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.19, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); BV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.74, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); BV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.79, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); BV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.11, ANOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.78, ANOVA
Statistical Analysis 7: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); OV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.90, ANOVA
Statistical Analysis 8: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); OV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.33, ANOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); OV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.51, ANOVA
Statistical Analysis 10: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); OV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.28, ANOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.86, ANOVA
Statistical Analysis 12: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); OS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.60, ANOVA
Statistical Analysis 13: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); OS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.84, ANOVA
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); OS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.98, ANOVA
Statistical Analysis 15: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); OS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.47, ANOVA
Statistical Analysis 16: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OcS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.59, ANOVA
Statistical Analysis 17: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); OcS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.13, ANOVA
Statistical Analysis 18: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); OcS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.65, ANOVA
Statistical Analysis 19: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); OcS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.33, ANOVA
Statistical Analysis 20: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); OcS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.053, ANOVA
Statistical Analysis 21: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); ObS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.51, ANOVA
Statistical Analysis 22: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); ObS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.50, ANOVA
Statistical Analysis 23: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); ObS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.27, ANOVA
Statistical Analysis 24: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); ObS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.091, ANOVA
Statistical Analysis 25: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); ObS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.087, ANOVA
Statistical Analysis 26: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); MS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.82, ANOVA
Statistical Analysis 27: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); MS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.82, ANOVA
Statistical Analysis 28: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); MS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.12, ANOVA
Statistical Analysis 29: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); MS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.085, ANOVA
Statistical Analysis 30: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); MS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.080, ANOVA
Statistical Analysis 31: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); ES: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.24, ANOVA
Statistical Analysis 32: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); ES: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.035, ANOVA
Statistical Analysis 33: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); ES: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.024, ANOVA
Statistical Analysis 34: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); ES: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.30, ANOVA
Statistical Analysis 35: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); ES: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.89, ANOVA
Statistical Analysis 36: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OMS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.80, ANOVA
Statistical Analysis 37: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); OMS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.75, ANOVA
Statistical Analysis 38: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); OMS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.060, ANOVA
Statistical Analysis 39: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); OMS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.12, ANOVA
Statistical Analysis 40: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); OMS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.13, ANOVA
Statistical Analysis 41: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); CP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.78, ANOVA
Statistical Analysis 42: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); CP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.70, ANOVA
Statistical Analysis 43: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); CP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.98, ANOVA
Statistical Analysis 44: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); CP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.76, ANOVA
Statistical Analysis 45: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); CP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.73, ANOVA

30. Secondary Outcome: Bone Histomorphometric Indices at Month 60: BV, OV, OS, OcS, ObS, MS, ES, OMS, CP
Description: as for outcome 29
Time Frame: Month 60
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Percentage of indices
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 3 | 5 | 1
Percentage of indices
  BV (n=2,4,1) | 20.315 (4.882) | 17.818 (3.452) | 21.590 (6.905)
  OV (n=2,4,1) | 2.550 (0.258) | 0.893 (0.183) | 2.790 (0.365)
  OS (n=2,4,1) | 20.270 (3.091) | 9.772 (2.186) | 23.870 (4.372)
  OcS (n=2,4,1) | 0.445 (0.137) | 0.173 (0.097) | 0.310 (0.193)
  ObS (n=2,4,1) | 7.170 (2.100) | 2.430 (1.485) | 7.260 (2.970)
  MS (n=2,4,1) | 6.910 (1.614) | 2.920 (1.142) | 9.780 (2.283)
  ES (n=2,4,1) | 1.225 (0.226) | 0.542 (0.160) | 0.990 (0.319)
  OMS (n=3,5,1) | 57.300 (21.483) | 43.060 (16.640) | 40.900 (37.209)
  CP (n=0,0,0) | NA (NA) — Data was not analyzed as there were not enough data points to perform the analyses. | NA (NA) — Data was not analyzed as there were not enough data points to perform the analyses. | NA (NA) — Data was not analyzed as there were not enough data points to perform the analyses.
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); BV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.70, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); BV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.65, ANOVA
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.006, ANOVA
Statistical Analysis 4: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); OV: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.010, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.050, ANOVA
Statistical Analysis 6: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); OS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.045, ANOVA
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OcS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.18, ANOVA
Statistical Analysis 8: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); OcS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.56, ANOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); ObS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.14, ANOVA
Statistical Analysis 10: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); ObS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.22, ANOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); MS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.11, ANOVA
Statistical Analysis 12: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); MS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.055, ANOVA
Statistical Analysis 13: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); ES: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.069, ANOVA
Statistical Analysis 14: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); ES: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.28, ANOVA
Statistical Analysis 15: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OMS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.62, ANOVA
Statistical Analysis 16: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); OMS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.96, ANOVA

31. Secondary Outcome: Bone Histomorphometric Indices at Month 36: WTh, OTh, TbTh, TbSp and CTh
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD. Calculated indices included: Wall Thickness (WTh), Osteoid Thickness (OTh), Trabecular Thickness (TbTh), Trabecular Separation (TbSp) and Cortical thickness (CTh). Trabecular separation defined as the thickness of the spaces as defined by binarization within the volume of interest.
Time Frame: Month 36
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: micrometer (mcm)
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 25 | 27 | 28 | 30
micrometer (mcm)
  WTh (n=25,27,28,30) | 31.348 (0.541) | 31.689 (0.521) | 31.089 (0.512) | 30.447 (0.494)
  OTh (n=25,27,28,30) | 6.180 (0.221) | 6.085 (0.212) | 5.554 (0.209) | 5.660 (0.202)
  TbTh (n=25,27,28,30) | 140.440 (7.128) | 146.296 (6.859) | 139.143 (6.735) | 131.333 (6.507)
  TbSp (n=25,27,28,30) | 865.040 (42.634) | 770.148 (41.024) | 880.571 (40.285) | 787.900 (38.919)
  CTh (n=25,27,27,30) | 891.480 (68.949) | 694.370 (66.346) | 781.593 (66.346) | 761.467 (62.941)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); WTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.22, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); WTh: p-value was calculated using ANOVA; Test type: Superiority or Other; p = 0.087, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); WTh: p-value was calculated using ANOVA; Test type: Superiority or Other; p = 0.37, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); WTh: p-value was calculated using ANOVA; Test type: Superiority or Other; p = 0.73, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); WTh: p-value was calculated using ANOVA; Test type: Superiority or Other; p = 0.41, ANOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.085, ANOVA
Statistical Analysis 7: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); OTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.15, ANOVA
Statistical Analysis 8: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); OTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.71, ANOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); OTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.042, ANOVA
Statistical Analysis 10: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); OTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.077, ANOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); TbTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.35, ANOVA
Statistical Analysis 12: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); TbTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.12, ANOVA
Statistical Analysis 13: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); TbTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.41, ANOVA
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); TbTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.90, ANOVA
Statistical Analysis 15: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); TbTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.46, ANOVA
Statistical Analysis 16: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); TbSp: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.18, ANOVA
Statistical Analysis 17: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); TbSp: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.75, ANOVA
Statistical Analysis 18: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); TbSp: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.10, ANOVA
Statistical Analysis 19: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); TbSp: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.79, ANOVA
Statistical Analysis 20: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); TbSp: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.057, ANOVA
Statistical Analysis 21: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); CTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.17, ANOVA
Statistical Analysis 22: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); CTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.46, ANOVA
Statistical Analysis 23: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); CTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.83, ANOVA
Statistical Analysis 24: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); CTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.25, ANOVA
Statistical Analysis 25: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); CTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.35, ANOVA

32. Secondary Outcome: Bone Histomorphometric Indices at Month 60: WTh, OTh, TbTh, TbSp and CTh
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD. Calculated indices included: WTh, OTh, TbTh, TbSp and CTh. Trabecular separation defined as the thickness of the spaces as defined by binarization within the volume of interest.
Time Frame: Month 60
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: mcm
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 2 | 4 | 1
mcm
  WTh (n=2,4,1) | 34.250 (0.833) | 30.300 (0.589) | 28.700 (1.177)
  OTh (n=2,4,1) | 7.450 (0.571) | 5.500 (0.404) | 6.400 (0.807)
  TbTh (n=2,4,1) | 154.500 (29.636) | 153.000 (20.956) | 139.000 (41.912)
  TbSp (n=2,4,1) | 748.000 (161.893) | 920.750 (114.476) | 628.000 (228.951)
  CTh (n=0,0,0) | NA (NA) — Data was not analyzed as there were not enough data points to perform the analyses. | NA (NA) — Data was not analyzed as there were not enough data points to perform the analyses. | NA (NA) — Data was not analyzed as there were not enough data points to perform the analyses.
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); WTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.018, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); WTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.29, ANOVA
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); OTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.049, ANOVA
Statistical Analysis 4: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); OTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.37, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); TbTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.97, ANOVA
Statistical Analysis 6: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); TbTh: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.78, ANOVA
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); TbSp: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.43, ANOVA
Statistical Analysis 8: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); TbSp: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.32, ANOVA

33. Secondary Outcome: Bone Histomorphometric Indices at Month 36: Total Surface (Goldner Slide) [TSG]
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD. Calculated indices included: Total Surface (Goldner Slide) [TSG]. All specimens were demineralized and subjected to staining procedures (Goldner's staining). Slides were analyzed using light microscopy for total surface area, the surface area that consisted of bone and the surface area that consisted of graft material (all in mm^2 and expressed as percent (%) of the total surface.
Time Frame: Month 36
Population: ITT population included all randomized participants who took at least 1 dose of test article; had baseline data and at least one valid bone histomorphometry while on therapy. 'N' (number of participants analyzed)=participants evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 28 | 29 | 32 | 32
millimeter (mm) | 95.111 (8.429) | 110.897 (8.283) | 94.353 (7.885) | 105.912 (7.885)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.35, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.66, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.30, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.95, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.15, ANOVA

34. Secondary Outcome: Bone Histomorphometric Indices at Month 60: TSG
Description: as for outcome 33
Time Frame: Month 60
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 3 | 5 | 1
mm | 75.333 (30.542) | 75.560 (23.658) | 128.500 (52.900)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 1.00, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.40, ANOVA

35. Secondary Outcome: Bone Histomorphometric Indices at Month 36: TtAr
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD. Calculated variable: Tissue Area (TtAr). Tissue area comprised of the porous calcified substance from which bones were made.
Time Frame: Month 36
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Square millimeter (mm^2)
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 28 | 29 | 32 | 32
Square millimeter (mm^2) | 39.904 (3.066) | 42.334 (3.013) | 39.497 (2.868) | 41.459 (2.868)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.71, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.83, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.63, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.92, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.50, ANOVA

36. Secondary Outcome: Bone Histomorphometric Indices at Month 60: TtAr
Description: as for outcome 35
Time Frame: Month 60
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 3 | 5 | 1
mm^2 | 28.767 (12.993) | 34.600 (10.064) | 41.200 (22.504)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.73, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.80, ANOVA

37. Secondary Outcome: Bone Histomorphometric Indices at Month 36: BFP, RP and RmP
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD. Calculated indices included: Bone Formation Period (BFP), Resorption Period (RP), Remodeling Period (RmP).
Time Frame: Month 36
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: years (yrs)
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 24 | 27 | 24 | 27
years (yrs)
  BFP (n=24,27,24,27) | 0.463 (0.080) | 0.441 (0.076) | 0.751 (0.080) | 0.436 (0.076)
  RP (n=24,27,24,27) | 0.080 (0.029) | 0.066 (0.027) | 0.125 (0.029) | 0.096 (0.027)
  RmP (n=24,27,24,27) | 0.543 (0.095) | 0.508 (0.090) | 0.876 (0.095) | 0.531 (0.090)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); BFP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.81, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); BFP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.96, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); BFP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.005, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); BFP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.013, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); BFP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.006, ANOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); RP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.70, ANOVA
Statistical Analysis 7: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); RP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.44, ANOVA
Statistical Analysis 8: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); RP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.47, ANOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); RP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.28, ANOVA
Statistical Analysis 10: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); RP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.14, ANOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); RmP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.93, ANOVA
Statistical Analysis 12: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); RmP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.85, ANOVA
Statistical Analysis 13: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); RmP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.010, ANOVA
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); RmP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.015, ANOVA
Statistical Analysis 15: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); RmP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.006, ANOVA

38. Secondary Outcome: Bone Histomorphometric Indices at Month 60: BFP, RP and RmP
Description: as for outcome 37
Time Frame: Month 60
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: yrs
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 2 | 4 | 1
yrs
  BFP (n=2,4,1) | 0.545 (0.391) | 0.820 (0.277) | 0.390 (0.553)
  RP (n=2,4,1) | 0.035 (0.011) | 0.035 (0.008) | 0.020 (0.015)
  RmP (n=2,4,1) | 0.580 (0.403) | 0.860 (0.285) | 0.410 (0.569)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); BFP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.60, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); BFP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.53, ANOVA
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); RP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 1.00, ANOVA
Statistical Analysis 4: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); RP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.43, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); RmP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.60, ANOVA
Statistical Analysis 6: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); RmP: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.52, ANOVA

39. Secondary Outcome: Bone Histomorphometric Indices at Month 36: SuD
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD Calculated indices included: Surface Density (SuD).
Time Frame: Month 36
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: square millimeter per cubic millimeter
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 25 | 27 | 28 | 30
square millimeter per cubic millimeter | 2.405 (0.109) | 2.632 (0.105) | 2.424 (0.103) | 2.587 (0.100)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.22, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.76, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.26, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.90, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.16, ANOVA

40. Secondary Outcome: Bone Histomorphometric Indices at Month 60: SuD
Description: as for outcome 39
Time Frame: Month 60
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: square millimeter per cubic millimeter
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 2 | 4 | 1
square millimeter per cubic millimeter | 2.625 (0.338) | 2.248 (0.239) | 3.120 (0.479)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.41, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.18, ANOVA

41. Secondary Outcome: Bone Histomorphometric Indices at Month 36: BFRTS
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD Calculated indices included: Bone Form Rate (BFR)-Total Surface Reference (BFRTS). BFR accounts the bone surface which is actively mineralizing, which depends on the number of osteoblasts that are active. BFR= Fraction of mineralizing surface and bone surface multiplied by mineralization apposition rate (MAR).
Time Frame: Month 36
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: cubic millimetre/square millimetre/year
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 24 | 27 | 24 | 27
cubic millimetre/square millimetre/year | 0.013 (0.002) | 0.012 (0.002) | 0.009 (0.002) | 0.012 (0.002)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.68, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.97, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.18, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.088, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.17, ANOVA

42. Secondary Outcome: Bone Histomorphometric Indices at Month 60: BFRTS
Description: as for outcome 41
Time Frame: Month 60
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: cubic millimetre/square millimetre/year
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 2 | 4 | 1
cubic millimetre/square millimetre/year | 0.013 (0.003) | 0.006 (0.002) | 0.018 (0.005)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.25, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.10, ANOVA

43. Secondary Outcome: Bone Histomorphometric Indices at Month 36: ACF
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD Calculated indices included: Activation Frequency (ACF). The total period (TP) is the duration between the beginning of one formation period (FP) and the beginning of the next FP. The number of times per year that this spot begins the FP is the activation frequency (ACF).
Time Frame: Month 36
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Activation of bone formation/year
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 24 | 27 | 24 | 27
Activation of bone formation/year | 0.421 (0.058) | 0.385 (0.054) | 0.290 (0.058) | 0.410 (0.054)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.90, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.74, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.13, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.11, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.24, ANOVA

44. Secondary Outcome: Bone Histomorphometric Indices at Month 60: ACF
Description: as for outcome 43
Time Frame: Month 60
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Activation of bone formation/year
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 2 | 4 | 1
Activation of bone formation/year | 0.375 (0.106) | 0.198 (0.075) | 0.610 (0.151)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.25, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.070, ANOVA

45. Secondary Outcome: Bone Histomorphometric Indices at Month 36: Mlt
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD Calculated indices included: Mineralization Lag Time (Mlt). Mineralization lag time was the lag between the time osteoid was formed and the mineral was added.
Time Frame: Month 36
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 24 | 27 | 24 | 27
days | 31.650 (5.141) | 30.337 (4.847) | 48.383 (5.141) | 29.533 (4.847)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.77, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.91, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.009, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.023, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.012, ANOVA

46. Secondary Outcome: Bone Histomorphometric Indices at Month 60: Mlt
Description: as for outcome 45
Time Frame: Month 60
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 2 | 4 | 1
days | 43.450 (21.817) | 51.100 (15.427) | 31.900 (30.855)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.79, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.61, ANOVA

47. Secondary Outcome: Bone Histomorphometric Indices at Month 36: MAR
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD Calculated indices included: Mineral Apposition Rate (MAR). MAR is the area of new bone formed during the label interval.
Time Frame: Month 36
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: mcm/days (mcm/d)
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 24 | 27 | 24 | 27
mcm/days (mcm/d) | 0.578 (0.020) | 0.563 (0.019) | 0.520 (0.020) | 0.550 (0.019)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.30, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.62, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.28, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.041, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.12, ANOVA

48. Secondary Outcome: Bone Histomorphometric Indices at Month 60: MAR
Description: as for outcome 47
Time Frame: Month 60
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: mcm/d
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 2 | 4 | 1
mcm/d | 0.525 (0.095) | 0.573 (0.067) | 0.490 (0.134)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.70, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.61, ANOVA

49. Secondary Outcome: Bone Histomorphometric Indices at Month 36: TbN
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD Calculated indices included: Trabecular Number (TbN). TbN= Ratio of bone volume to tissue volume divided by trabecular thickness.
Time Frame: Month 36
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: ratio/millimeter (ratio/mm)
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 25 | 27 | 28 | 30
ratio/millimeter (ratio/mm) | 1.202 (0.055) | 1.315 (0.053) | 1.212 (0.052) | 1.293 (0.050)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.22, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.76, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.26, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.89, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.17, ANOVA

50. Secondary Outcome: Bone Histomorphometric Indices at Month 60: TbN
Description: as for outcome 49
Time Frame: Month 60
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: ratio/mm
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 2 | 4 | 1
ratio/mm | 1.315 (0.168) | 1.125 (0.119) | 1.560 (0.238)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.41, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.18, ANOVA

51. Secondary Outcome: Bone Histomorphometric Indices at Month 36: BFRBV
Description: Bone histomorphometry verified rate of bone remodeling. Anterior iliac crest bone biopsy done to exclude presence of osteomalacia or more subtle defects in mineralization; investigated qualitative aspects of bone. Also assessed decrease in rate of bone turnover, investigated mechanism for observed increase in BMD Calculated indices included: Bone Formation Rate (BFR)-Bone Volume Reference (BFRBV). BFR accounts the bone volume which is actively mineralizing, which depends on the number of osteoblasts that are active. BFR= Fraction of mineralizing volume and bone volume multiplied by mineralization apposition rate (MAR).
Time Frame: Month 36
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: square millimetre/square millimetre/year
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 24 | 27 | 24 | 27
square millimetre/square millimetre/year | 0.186 (0.024) | 0.171 (0.022) | 0.122 (0.024) | 0.187 (0.022)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.97, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.61, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.050, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.061, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Test type: Superiority or Other; p = 0.14, ANOVA

52. Secondary Outcome: Bone Histomorphometric Indices at Month 60: BFRBV
Description: as for outcome 51
Time Frame: Month 60
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: square millimetre/square millimetre/year
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Placebo (Core+SE I+SE II) | Bazedoxifene 40/20 mg (SE I)
Number analyzed (Participants) | 2 | 4 | 1
square millimetre/square millimetre/year | 0.167 (0.042) | 0.075 (0.030) | 0.253 (0.059)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Test type: Superiority or Other; p = 0.15, ANOVA
Statistical Analysis 2: Comparison: Placebo (Core+SE I+SE II) vs Bazedoxifene 40/20 mg (SE I); Test type: Superiority or Other; p = 0.056, ANOVA

53. Secondary Outcome: Women's Health Questionnaire (WHQ)
Description: WHQ is a measure of mid-aged women's emotional and physical health. Consists of 36-item assessing nine domains of physical and emotional health: Depressed mood; Somatic symptoms; Anxiety/fears; Vasomotor symptoms; Sleep problems; Sexual behavior; Menstrual symptoms; Memory/concentration; and Attractiveness. Each item scored on a 4 point scale (yes definitely, yes sometimes, not much, no not at all) reduced to binary option as 0 (no) and 1 (yes). Domain subscale score was calculated as sum of domain items score divided by number of domain items. Total score was calculated as the sum of individual domain subscale score divided by number of domains. Total score range from 0 (absent) to 1 (present), with higher scores indicating more pronounced distress and dysfunction. Baseline values at different time points were considered only for the participants who were evaluable at those time points.
Time Frame: Baseline
Population: ITT population included all randomized participants who took at least 1 dose of test article;had baseline data and at least one valid assessment while on therapy. 'N' (number of participants analyzed)=participants evaluable for this measure. 'n'=participants who were evaluable for this measure at the specified time point for each arm group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1490 | 1435 | 1461 | 1503
Units on a scale
  Baseline: Month 12 (n=1490,1435,1461,1503) | 0.342 (0.176) | 0.348 (0.176) | 0.341 (0.182) | 0.343 (0.182)
  Baseline: Month 24 (n=1307,1271,1311,1318) | 0.339 (0.175) | 0.343 (0.176) | 0.338 (0.183) | 0.343 (0.181)
  Baseline: Month 36 (n=1153,1138,1168,1179) | 0.333 (0.173) | 0.341 (0.175) | 0.341 (0.182) | 0.339 (0.180)

54. Secondary Outcome: Change From Baseline in Women's Health Questionnaire (WHQ) at Month 12, 24 and 36
Description: WHQ is a measure of mid-aged women's emotional and physical health. Consists of 36-item assessing nine domains of physical and emotional health: Depressed mood; Somatic symptoms; Anxiety/fears; Vasomotor symptoms; Sleep problems; Sexual behavior; Menstrual symptoms; Memory/concentration; and Attractiveness. Each item scored on a 4 point scale (yes definitely, yes sometimes, not much, no not at all) reduced to binary option as 0 (no) and 1 (yes). Domain subscale score was calculated as sum of domain items score divided by number of domain items. Total score was calculated as the sum of individual domain subscale score divided by number of domains. Total score range from 0 (absent) to 1 (present), with higher scores indicating more pronounced distress and dysfunction.Baseline values at different time points were considered only for the participants who were evaluable at those time points.
Time Frame: Baseline, Months 12, 24, 36
Population: as for outcome 53
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1409 | 1435 | 1461 | 1503
Units on a scale
  Change at Month 12 (n=1490,1435,1461,1503) | 0.000 (0.003) | 0.001 (0.003) | 0.001 (0.003) | -0.005 (0.003)
  Change at Month 24 (n=1307,1271,1311,1318) | 0.005 (0.004) | 0.006 (0.004) | 0.007 (0.004) | -0.002 (0.004)
  Change at Month 36 (n=1153,1138,1168,1179) | 0.011 (0.005) | -0.000 (0.005) | 0.005 (0.005) | 0.005 (0.005)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 12 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.20, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 12 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.12, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 12 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.17, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 12 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.92, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 12 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.86, ANOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 24 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.18, ANOVA
Statistical Analysis 7: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 24 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.12, ANOVA
Statistical Analysis 8: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 24 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.096, ANOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 24 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.76, ANOVA
Statistical Analysis 10: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 24 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.93, ANOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 36 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.36, ANOVA
Statistical Analysis 12: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 36 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.34, ANOVA
Statistical Analysis 13: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 36 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.98, ANOVA
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 36 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.35, ANOVA
Statistical Analysis 15: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 36 in WHQ: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.35, ANOVA

55. Secondary Outcome: European Foundation for Osteoporosis Quality of Life Questionnaire (QUALEFFO)
Description: QUALEFFO is an osteoporosis-specific health instrument developed specifically for participants with vertebral deformities used to evaluate the effect of back pain and treatment on quality of life. The QUALEFFO questionnaire includes 41 items in 5 domains: pain, physical function, social function, general health perception, and mental function. The total score is calculated according to the scoring algorithm developed by the International Osteoporosis Foundation. Total scores are reported from 0 to 100, with lower scores corresponding to better quality of life. Baseline values at different time points were considered only for the participants who were evaluable at those time points.
Time Frame: Baseline
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1490 | 1438 | 1455 | 1495
Units on a scale
  Baseline: Month 12 (n=1490,1438,1455,1495) | 24.57 (12.95) | 24.50 (12.70) | 23.98 (12.54) | 24.31 (12.62)
  Baseline: Month 24 (n=1305,1276,1307,1312) | 24.33 (12.75) | 24.24 (12.58) | 23.80 (12.62) | 24.29 (12.60)
  Baseline: Month 36 (n=1155,1136,1168,1176) | 23.87 (12.70) | 24.12 (12.42) | 23.88 (12.51) | 23.97 (12.27)

56. Secondary Outcome: Change From Baseline in European Foundation for Osteoporosis Quality of Life Questionnaire (QUALEFFO) at Month 12, 24 and 36
Description: as for outcome 55
Time Frame: Baseline, Months 12, 24, 36
Population: as for outcome 53
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1490 | 1438 | 1455 | 1495
Units on a scale
  Change at Month 12 (n=1490,1438,1455,1495) | -0.24 (0.23) | -0.91 (0.24) | -0.49 (0.24) | -0.77 (0.23)
  Change at Month 24 (n=1305,1276,1307,1312) | -0.00 (0.27) | 0.02 (0.28) | 0.29 (0.27) | -0.39 (0.27)
  Change at Month 36 (n=1155,1136,1168,1176) | 0.62 (0.30) | -0.11 (0.30) | 0.26 (0.30) | -0.35 (0.30)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 12 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.080, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 12 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.41, ANOVA
Statistical Analysis 3: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 12 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.65, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 12 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.18, ANOVA
Statistical Analysis 5: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 12 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.36, ANOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 24 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.27, ANOVA
Statistical Analysis 7: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 24 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.25, ANOVA
Statistical Analysis 8: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 24 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.053, ANOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 24 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.40, ANOVA
Statistical Analysis 10: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 24 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.45, ANOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 36 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.012, ANOVA
Statistical Analysis 12: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 36 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.54, ANOVA
Statistical Analysis 13: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 36 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.11, ANOVA
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 36 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.35, ANOVA
Statistical Analysis 15: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 36 in QUALEFFO: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.34, ANOVA

57. Secondary Outcome: Euro Quality of Life-5 Dimensions (EQ-5D) Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state. Baseline values at different time points were considered only for the participants who were evaluable at those time points.
Time Frame: Baseline
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1381 | 1346 | 1362 | 1407
millimeter (mm)
  Baseline: Month 12 (n=1381,1346,1362,1407) | 79.20 (18.05) | 80.89 (39.47) | 82.23 (45.23) | 80.95 (32.47)
  Baseline: Month 24 (n=1210,1200,1223,1247) | 79.11 (17.99) | 80.73 (33.66) | 82.86 (49.89) | 80.79 (31.66)
  Baseline: Month 36 (n=1070,1065,1092,1120) | 79.78 (18.00) | 81.43 (35.02) | 83.50 (52.36) | 81.07 (31.54)

58. Secondary Outcome: Change From Baseline in Euro Quality of Life-5 Dimensions (EQ-5D) Visual Analog Scale (VAS) at Month 12, 24 and 36
Description: as for outcome 57
Time Frame: Baseline, Months 12, 24, 36
Population: as for outcome 53
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1381 | 1346 | 1362 | 1407
mm
  Change at Month 12 (n=1381,1346,1362,1407) | 1.59 (1.23) | 0.12 (1.24) | -1.39 (1.23) | -0.37 (1.21)
  Change at Month 24 (n=1210,1200,1223,1247) | 0.45 (1.39) | -1.13 (1.40) | -1.63 (1.37) | -2.12 (1.37)
  Change at Month 36 (n=1070,1065,1092,1120) | 5.73 (1.74) | 3.87 (1.74) | 1.60 (1.71) | 4.66 (1.70)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 12 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.21, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 12 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.058, ANOVA
Statistical Analysis 3: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 12 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.76, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 12 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.34, ANOVA
Statistical Analysis 5: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 12 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.51, ANOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 24 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.14, ANOVA
Statistical Analysis 7: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 24 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.57, ANOVA
Statistical Analysis 8: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 24 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.78, ANOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 24 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.24, ANOVA
Statistical Analysis 10: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 24 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.78, ANOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 36 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.62, ANOVA
Statistical Analysis 12: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 36 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.72, ANOVA
Statistical Analysis 13: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 36 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.16, ANOVA
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 36 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.059, ANOVA
Statistical Analysis 15: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 36 in EQ-5D VAS: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.30, ANOVA

59. Secondary Outcome: Euro Quality of Life-5 Dimensions (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. Baseline values at different time points were considered only for the participants who were evaluable at those time points.
Time Frame: Baseline
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1425 | 1375 | 1393 | 1436
Units on a scale
  Baseline: Month 12 (n=1425,1375,1393,1436) | 0.81 (0.20) | 0.82 (0.20) | 0.82 (0.19) | 0.81 (0.21)
  Baseline: Month 24 (n=1243,1220,1240,1267) | 0.81 (0.20) | 0.82 (0.19) | 0.82 (0.19) | 0.81 (0.21)
  Baseline: Month 36 (n=1095,1078,1111,1128) | 0.82 (0.20) | 0.82 (0.18) | 0.82 (0.19) | 0.82 (0.20)

60. Secondary Outcome: Change From Baseline in Euro Quality of Life-5 Dimensions (EQ-5D)- Health State Profile Utility Score at Month 12, 24 and 36
Description: as for outcome 59
Time Frame: Baseline, Months 12, 24, 36
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bazedoxifene 20 mg (Core+SE I) | Bazedoxifene 40 mg (Core) | Raloxifene 60 mg (Core) | Placebo (Core+SE I+SE II)
Number analyzed (Participants) | 1425 | 1375 | 1393 | 1436
Units on a scale
  Change at Month 12 (n=1425,1375,1393,1436) | 0.01 (0.01) | 0.01 (0.01) | 0.01 (0.01) | 0.01 (0.01)
  Change at Month 24(n=1243,1220,1240,1267) | 0.00 (0.01) | -0.01 (0.01) | -0.01 (0.01) | 0.01 (0.01)
  Change at Month 36 (n=1095,1078,1111,1128) | -0.00 (0.01) | -0.01 (0.01) | -0.01 (0.01) | -0.00 (0.01)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 12 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.72, ANOVA
Statistical Analysis 2: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 12 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.98, ANOVA
Statistical Analysis 3: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 12 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.84, ANOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 12 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.88, ANOVA
Statistical Analysis 5: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 12 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.86, ANOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 24 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.82, ANOVA
Statistical Analysis 7: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 24 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.11, ANOVA
Statistical Analysis 8: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 24 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.14, ANOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 24 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.22, ANOVA
Statistical Analysis 10: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 24 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.88, ANOVA
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Placebo (Core+SE I+SE II); Change at Month 36 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.96, ANOVA
Statistical Analysis 12: Comparison: Bazedoxifene 40 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 36 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.76, ANOVA
Statistical Analysis 13: Comparison: Raloxifene 60 mg (Core) vs Placebo (Core+SE I+SE II); Change at Month 36 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.92, ANOVA
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg (Core+SE I) vs Raloxifene 60 mg (Core); Change at Month 36 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.89, ANOVA
Statistical Analysis 15: Comparison: Bazedoxifene 40 mg (Core) vs Raloxifene 60 mg (Core); Change at Month 36 in EQ-5D: P value was calculated using ANOVA; Test type: Superiority or Other; p = 0.83, ANOVA

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Bazedoxifene 20 mg: Bazedoxifene acetate 20 mg capsule orally once daily along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily in core study, study extension I and II.
- Bazedoxifene 40/ 20 mg: Bazedoxifene acetate 40 mg capsule orally once daily in the core study, in first year of study extension I and then dose reduced to bazedoxifene acetate 20 mg in second year of study extension I, and II along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily.
- Raloxifene 60 mg (Core Study): Raloxifene 60 mg capsule orally once daily in the core study along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily.
- Placebo: Matching placebo capsule orally once daily along with supplement tablet (containing calcium up to 600 mg and vitamin D up to 400 IU) orally twice daily in the core study, study extension I and II.
Arm/Group | Bazedoxifene 20 mg | Bazedoxifene 40/ 20 mg | Raloxifene 60 mg (Core Study) | Placebo
Serious Adverse Events (participants affected / at risk) | 507/1886 | 468/1872 | 393/1849 | 479/1885
Other Adverse Events (participants affected / at risk) | 1818/1886 | 1800/1872 | 1775/1849 | 1823/1885
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bazedoxifene 20 mg (N=1886) | Bazedoxifene 40/ 20 mg (N=1872) | Raloxifene 60 mg (Core Study) (N=1849) | Placebo (N=1885)
Abdominal pain (General disorders) | 7 | 6 | 8 | 8
Abdominal syndrome acute (General disorders) | 4 | 9 | 5 | 5
Abscess (General disorders) | 8 | 2 | 3 | 3
Accidental injury (General disorders) | 65 | 50 | 55 | 61
Accidental overdose (General disorders) | 4 | 4 | 5 | 3
Adenoma (General disorders) | 1 | 2 | 1 | 2
Allergic reaction (General disorders) | 0 | 2 | 1 | 1
Anaphylactoid reaction (General disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 2 | 0 | 3
Back pain (General disorders) | 9 | 4 | 6 | 4
Carcinoma (General disorders) | 6 | 5 | 2 | 2
Cellulitis (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 6 | 9 | 10 | 12
Chest pain substernal (General disorders) | 3 | 4 | 0 | 3
Collagen disorder (General disorders) | 1 | 0 | 0 | 0
Cyst (General disorders) | 6 | 0 | 1 | 0
Death (General disorders) | 0 | 3 | 0 | 1
Fever (General disorders) | 2 | 1 | 1 | 4
Fibrosis (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Headache (General disorders) | 0 | 0 | 1 | 1
Hernia (General disorders) | 9 | 6 | 9 | 12
Human immunodeficiency virus test positive (General disorders) | 1 | 0 | 0 | 1
Hormone level altered (General disorders) | 0 | 0 | 0 | 1
Hydrocephalus (General disorders) | 0 | 0 | 0 | 1
Hyperplasia (General disorders) | 0 | 0 | 0 | 1
Infection (General disorders) | 6 | 10 | 10 | 10
Lab test abnormal (General disorders) | 1 | 0 | 1 | 0
Malaise (General disorders) | 1 | 1 | 1 | 0
Neck pain (General disorders) | 2 | 1 | 0 | 0
Neoplasm (General disorders) | 8 | 6 | 3 | 9
Non-specified drug reaction (General disorders) | 1 | 0 | 0 | 0
Overdose (General disorders) | 10 | 8 | 10 | 10
Pain (General disorders) | 2 | 3 | 5 | 2
Peritonitis (General disorders) | 3 | 1 | 1 | 2
Sarcoma (General disorders) | 0 | 2 | 0 | 1
Sepsis (General disorders) | 3 | 1 | 2 | 3
Septic shock (General disorders) | 4 | 0 | 1 | 1
Suicide attempt (General disorders) | 0 | 1 | 0 | 0
Aneurysm (Cardiac disorders) | 0 | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 13 | 6 | 10 | 9
Aortic stenosis (Cardiac disorders) | 3 | 4 | 2 | 2
Arrhythmia (Cardiac disorders) | 4 | 1 | 2 | 0
Arterial anomaly (Cardiac disorders) | 1 | 1 | 0 | 2
Arterial thrombosis (Cardiac disorders) | 1 | 1 | 0 | 0
Arteriosclerosis (Cardiac disorders) | 1 | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 9 | 10 | 6 | 6
Atrial flutter (Cardiac disorders) | 2 | 1 | 0 | 0
AV block (Cardiac disorders) | 1 | 1 | 1 | 0
AV block complete (Cardiac disorders) | 0 | 0 | 0 | 1
AV block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 2 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 2 | 1 | 1
Carotid occlusion (Cardiac disorders) | 0 | 0 | 0 | 1
Carotid thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0
Cerebral hemorrhage (Cardiac disorders) | 1 | 1 | 0 | 2
Cerebral infarct (Cardiac disorders) | 0 | 4 | 1 | 2
Cerebral ischemia (Cardiac disorders) | 6 | 10 | 6 | 7
Cerebral thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Cardiac disorders) | 14 | 17 | 10 | 18
Cerebrovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 1
Congestive heart failure (Cardiac disorders) | 3 | 4 | 3 | 2
Coronary artery disorder (Cardiac disorders) | 9 | 8 | 5 | 3
Coronary occlusion (Cardiac disorders) | 1 | 1 | 0 | 1
Deep vein thrombosis (Cardiac disorders) | 8 | 13 | 10 | 3
Electrocardiogram abnormal (Cardiac disorders) | 0 | 0 | 2 | 0
Embolus lower extremity (Cardiac disorders) | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Heart arrest (Cardiac disorders) | 0 | 0 | 1 | 4
Heart block (Cardiac disorders) | 0 | 0 | 1 | 0
Heart failure (Cardiac disorders) | 3 | 5 | 6 | 1
Hemorrhage (Cardiac disorders) | 0 | 0 | 2 | 0
Hypertension (Cardiac disorders) | 13 | 8 | 18 | 17
Hypertensive encephalopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Hypotension (Cardiac disorders) | 0 | 0 | 1 | 0
Infarct (Cardiac disorders) | 0 | 0 | 1 | 0
Intracranial aneurysm (Cardiac disorders) | 0 | 1 | 2 | 0
Intracranial hemorrhage (Cardiac disorders) | 0 | 1 | 1 | 1
Mesenteric occlusion (Cardiac disorders) | 0 | 0 | 1 | 0
Migraine (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarct (Cardiac disorders) | 9 | 10 | 8 | 11
Myocardial ischemia (Cardiac disorders) | 6 | 1 | 3 | 1
Palpitation (Cardiac disorders) | 2 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 1 | 0 | 0
Peripheral gangrene (Cardiac disorders) | 0 | 1 | 0 | 0
Peripheral vascular disorder (Cardiac disorders) | 3 | 1 | 1 | 0
Phlebitis (Cardiac disorders) | 0 | 0 | 0 | 1
Pulmonary embolus (Cardiac disorders) | 7 | 3 | 4 | 4
Pulmonary hypertension (Cardiac disorders) | 0 | 0 | 0 | 1
Retinal artery occlusion (Cardiac disorders) | 1 | 0 | 1 | 1
Retinal vein thrombosis (Cardiac disorders) | 0 | 2 | 1 | 2
Shock (Cardiac disorders) | 3 | 3 | 2 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 2 | 1 | 1
Subarachnoid hemorrhage (Cardiac disorders) | 0 | 2 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 3 | 1 | 0 | 2
Syncope (Cardiac disorders) | 8 | 9 | 4 | 6
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 1
Tachycardia sinus (Cardiac disorders) | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Cardiac disorders) | 4 | 6 | 3 | 0
Thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0
Valvular heart disease (Cardiac disorders) | 3 | 1 | 2 | 0
Varicose vein (Cardiac disorders) | 8 | 2 | 3 | 5
Vascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0
Vascular purpura (Cardiac disorders) | 1 | 0 | 0 | 0
Vasculitis (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Biliary pain (Gastrointestinal disorders) | 2 | 2 | 3 | 1
Blood in stool (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Carcinoma of mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholangitis (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Cholecystitis (Gastrointestinal disorders) | 12 | 12 | 6 | 11
Cholelithiasis (Gastrointestinal disorders) | 21 | 23 | 13 | 31
Cholestatic jaundice (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Cleft palate (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 5 | 9 | 1 | 6
Constipation (Gastrointestinal disorders) | 6 | 4 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 3
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Esophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fecal impaction (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 4 | 1 | 2 | 2
Gastroenteritis (Gastrointestinal disorders) | 2 | 1 | 2 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 4
Gastrointestinal carcinoma (Gastrointestinal disorders) | 15 | 13 | 11 | 17
Gastrointestinal disorder (Gastrointestinal disorders) | 5 | 2 | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 | 1 | 1 | 3
GI neoplasia (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hemorrhage of colon (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hemorrhagic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hemorrhagic pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hepatic neoplasia (Gastrointestinal disorders) | 0 | 3 | 2 | 0
Hepatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatomegaly (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatal hernia (Gastrointestinal disorders) | 3 | 2 | 1 | 2
Ileitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 3 | 2 | 3
Intestinal obstruction (Gastrointestinal disorders) | 4 | 1 | 1 | 4
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Jaundice (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Liver damage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Liver function tests abnormal (Gastrointestinal disorders) | 3 | 3 | 1 | 7
Malabsorption syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Megacolon (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 3
Pancreas disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 2 | 3 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyloric stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal disorder (Gastrointestinal disorders) | 11 | 7 | 1 | 7
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Sialadenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomach ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 5
Stomach ulcer hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ulcerative colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2 | 7
Adh inappropriate (Endocrine disorders) | 1 | 0 | 0 | 0
Diabetes mellitus (Endocrine disorders) | 2 | 5 | 1 | 1
Goiter (Endocrine disorders) | 4 | 5 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Parathyroid disorder (Endocrine disorders) | 1 | 0 | 0 | 4
Thyroid adenoma (Endocrine disorders) | 2 | 1 | 1 | 0
Thyroid carcinoma (Endocrine disorders) | 5 | 0 | 0 | 1
Thyroid disorder (Endocrine disorders) | 0 | 3 | 2 | 1
Thyroid neoplasia (Endocrine disorders) | 0 | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0
Acute myeloblastic leukemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 4
Chronic lymphocytic leukemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Ecchymosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
Lymphoma (Blood and lymphatic system disorders) | 1 | 1 | 2 | 4
Lymphoma like reaction (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Myeloma (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Myeloproliferative disorder (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Petechiae (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4
Bilirubinemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 3 | 5
Edema (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Electrolyte abnormality (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Healing abnormal (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1
Hypercholesteremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperlipemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Peripheral edema (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Serum glutamic oxaloacetic transaminase increased (Metabolism and nutrition disorders) | 1 | 1 | 0 | 5
Serum glutamic pyruvic transaminase increased (Metabolism and nutrition disorders) | 2 | 1 | 1 | 7
Weight gain (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Weight loss (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 7 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 7 | 4 | 0 | 4
Arthrosis (Musculoskeletal and connective tissue disorders) | 26 | 25 | 22 | 23
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Chondrodystrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Meniscus lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal anomaly (Musculoskeletal and connective tissue disorders) | 3 | 9 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Myasthenia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendon rupture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Addiction (Nervous system disorders) | 1 | 0 | 0 | 0
Alcoholism (Nervous system disorders) | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 3 | 1 | 0 | 0
Anxiety (Nervous system disorders) | 1 | 0 | 1 | 3
Apathy (Nervous system disorders) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Central nervous system neoplasia (Nervous system disorders) | 0 | 2 | 3 | 1
Confusion (Nervous system disorders) | 0 | 2 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Nervous system disorders) | 3 | 3 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 5
Emotional lability (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Extrapyramidal syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0
Hallucinations (Nervous system disorders) | 0 | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 1 | 0 | 1
Hypesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Manic depressive reaction (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Mental status changes (Nervous system disorders) | 0 | 0 | 2 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 2
Neuralgia (Nervous system disorders) | 2 | 0 | 2 | 0
Neuritis (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0
Ophthalmoplegia (Nervous system disorders) | 0 | 0 | 1 | 0
Paralysis (Nervous system disorders) | 0 | 1 | 1 | 0
Paresis (Nervous system disorders) | 3 | 1 | 1 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 3 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0
Personality disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Radiculopathy nos (Nervous system disorders) | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Subdural hematoma (Nervous system disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Nervous system disorders) | 1 | 0 | 0 | 0
Suicide (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 4 | 1 | 0 | 2
Vertigo (Nervous system disorders) | 1 | 2 | 2 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 3
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 4 | 3
Carcinoma of lung (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 5 | 5
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 5 | 7
Cough increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal neoplasia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 2
Lung edema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 21 | 19 | 15 | 23
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Discoid lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Fungal dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin benign neoplasm (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin carcinoma (Skin and subcutaneous tissue disorders) | 18 | 33 | 14 | 23
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin melanoma (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 3
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Sweating (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Abnormal vision (General disorders) | 1 | 0 | 1 | 1
Blindness transient (General disorders) | 1 | 2 | 0 | 0
Cataract specified (General disorders) | 7 | 2 | 4 | 1
Deafness (General disorders) | 0 | 1 | 2 | 0
Ear disorder (General disorders) | 0 | 0 | 0 | 2
Eye disorder (General disorders) | 0 | 2 | 0 | 0
Eye hemorrhage (General disorders) | 1 | 0 | 0 | 0
Glaucoma (General disorders) | 2 | 1 | 1 | 0
Keratitis (General disorders) | 0 | 1 | 0 | 0
Ophthalmitis (General disorders) | 1 | 0 | 0 | 0
Optic neuritis (General disorders) | 1 | 0 | 0 | 0
Otitis media (General disorders) | 0 | 1 | 0 | 0
Retinal degeneration (General disorders) | 0 | 1 | 0 | 2
Retinal detachment (General disorders) | 1 | 1 | 1 | 0
Retinal disorder (General disorders) | 2 | 1 | 1 | 1
Tinnitus (General disorders) | 0 | 1 | 0 | 0
Vestibular disorder (General disorders) | 0 | 1 | 1 | 0
Vitreous disorder (General disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Acute kidney failure (Renal and urinary disorders) | 1 | 0 | 0 | 1
Anuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bladder carcinoma (Renal and urinary disorders) | 2 | 2 | 2 | 1
Bladder neoplasm (Renal and urinary disorders) | 0 | 1 | 1 | 1
Breast carcinoma (Renal and urinary disorders) | 14 | 9 | 9 | 11
Breast cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast disorder (Renal and urinary disorders) | 1 | 3 | 0 | 0
Breast enlargement (Renal and urinary disorders) | 0 | 0 | 1 | 0
Breast neoplasm (Renal and urinary disorders) | 1 | 5 | 1 | 2
Cervix carcinoma (Renal and urinary disorders) | 0 | 1 | 3 | 0
Cervix carcinoma in situ (Renal and urinary disorders) | 2 | 0 | 0 | 0
Cervix disorder (Renal and urinary disorders) | 1 | 1 | 2 | 2
Cervix neoplasm (Renal and urinary disorders) | 2 | 1 | 2 | 3
Cystitis (Renal and urinary disorders) | 0 | 4 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Endometrial carcinoma (Renal and urinary disorders) | 0 | 3 | 2 | 7
Endometrial disorder (Renal and urinary disorders) | 2 | 1 | 1 | 1
Endometrial hyperplasia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Endometrial neoplasia (Renal and urinary disorders) | 5 | 4 | 3 | 6
Genital leukoplakia (Renal and urinary disorders) | 1 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 3 | 0 | 0
Kidney calculus (Renal and urinary disorders) | 4 | 1 | 0 | 2
Kidney failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Kidney function abnormal (Renal and urinary disorders) | 1 | 1 | 1 | 1
Ovarian carcinoma (Renal and urinary disorders) | 5 | 1 | 4 | 0
Ovarian cyst (Renal and urinary disorders) | 4 | 1 | 3 | 5
Ovarian disorder (Renal and urinary disorders) | 3 | 1 | 2 | 1
Ovarian germ cell teratoma benign (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pyelonephritis (Renal and urinary disorders) | 7 | 3 | 1 | 3
Urinary incontinence (Renal and urinary disorders) | 6 | 4 | 7 | 9
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 9 | 9 | 8 | 8
Urinary tract infection (Renal and urinary disorders) | 6 | 2 | 2 | 3
Urination impaired (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urogenital anomaly (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urogenital disorder (Renal and urinary disorders) | 1 | 0 | 1 | 1
Urolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Uterine disorder (Renal and urinary disorders) | 7 | 10 | 7 | 9
Uterine fibroids enlarged (Renal and urinary disorders) | 1 | 0 | 2 | 2
Vaginitis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vulvovaginal disorder (Renal and urinary disorders) | 2 | 1 | 1 | 5
Reaction unevaluable (General disorders) | 0 | 0 | 2 | 0
Adverse event associated with miscellaneous factors (General disorders) | 6 | 4 | 4 | 5
Allergic reaction other than drug (General disorders) | 0 | 0 | 1 | 0
Device malfunction (General disorders) | 0 | 0 | 3 | 0
Local reaction to procedure (Skin and subcutaneous tissue disorders) | 5 | 3 | 0 | 3
Surgical procedure (Surgical and medical procedures) | 1 | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bazedoxifene 20 mg (N=1886) | Bazedoxifene 40/ 20 mg (N=1872) | Raloxifene 60 mg (Core Study) (N=1849) | Placebo (N=1885)
Abdominal pain (General disorders) | 460 | 460 | 460 | 509
Accidental injury (General disorders) | 503 | 449 | 406 | 522
Asthenia (General disorders) | 234 | 230 | 220 | 226
Back pain (General disorders) | 676 | 652 | 632 | 674
Chest pain (General disorders) | 181 | 170 | 156 | 156
Flu syndrome (General disorders) | 536 | 523 | 529 | 559
Headache (General disorders) | 469 | 468 | 427 | 471
Infection (General disorders) | 526 | 514 | 462 | 516
Neck pain (General disorders) | 176 | 174 | 153 | 188
Pain (General disorders) | 643 | 616 | 615 | 659
Hypertension (Cardiac disorders) | 495 | 482 | 412 | 475
Vasodilatation (Cardiac disorders) | 247 | 253 | 227 | 127
Anorexia (Gastrointestinal disorders) | 80 | 72 | 100 | 97
Constipation (Gastrointestinal disorders) | 383 | 373 | 344 | 358
Diarrhea (Gastrointestinal disorders) | 196 | 237 | 221 | 217
Dyspepsia (Gastrointestinal disorders) | 215 | 202 | 185 | 223
Gastritis (Gastrointestinal disorders) | 127 | 106 | 100 | 93
Gastroenteritis (Gastrointestinal disorders) | 93 | 103 | 80 | 96
Nausea (Gastrointestinal disorders) | 177 | 176 | 158 | 176
Vomiting (Gastrointestinal disorders) | 120 | 118 | 119 | 137
Hypercholesteremia (Metabolism and nutrition disorders) | 211 | 162 | 115 | 231
Hyperglycemia (Metabolism and nutrition disorders) | 118 | 102 | 82 | 131
Hyperlipemia (Metabolism and nutrition disorders) | 139 | 125 | 97 | 133
Peripheral edema (Metabolism and nutrition disorders) | 239 | 217 | 208 | 192
Arthralgia (Musculoskeletal and connective tissue disorders) | 679 | 660 | 643 | 662
Arthrosis (Musculoskeletal and connective tissue disorders) | 192 | 200 | 172 | 200
Leg cramps (Musculoskeletal and connective tissue disorders) | 265 | 264 | 240 | 204
Myalgia (Musculoskeletal and connective tissue disorders) | 102 | 90 | 116 | 114
Anxiety (Nervous system disorders) | 101 | 106 | 108 | 137
Depression (Nervous system disorders) | 142 | 158 | 124 | 131
Dizziness (Nervous system disorders) | 232 | 198 | 176 | 212
Insomnia (Nervous system disorders) | 193 | 173 | 166 | 202
Paresthesia (Nervous system disorders) | 103 | 110 | 83 | 108
Vertigo (Nervous system disorders) | 171 | 141 | 149 | 167
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 209 | 218 | 158 | 193
Cough increased (Respiratory, thoracic and mediastinal disorders) | 251 | 231 | 192 | 234
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 171 | 192 | 166 | 213
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 87 | 91 | 83 | 103
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 125 | 119 | 111 | 112
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 167 | 156 | 127 | 151
Pruritus (Skin and subcutaneous tissue disorders) | 144 | 139 | 129 | 143
Rash (Skin and subcutaneous tissue disorders) | 85 | 87 | 79 | 98
Cataract specified (General disorders) | 119 | 121 | 91 | 126
Breast disorder (Renal and urinary disorders) | 135 | 137 | 109 | 153
Cervix disorder (Renal and urinary disorders) | 138 | 174 | 146 | 183
Cystitis (Renal and urinary disorders) | 111 | 121 | 106 | 102
Dysuria (Renal and urinary disorders) | 88 | 95 | 80 | 89
Urinary tract infection (Renal and urinary disorders) | 223 | 214 | 209 | 211
Vaginitis (Renal and urinary disorders) | 117 | 111 | 102 | 143
Adverse event associated with miscellaneous factors (General disorders) | 111 | 86 | 92 | 115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.